CLINICAL TRIAL: NCT02564055
Title: Study 203121: A Randomized, Blinded, Vehicle-Controlled, Dose-Finding Study of GSK2894512 Cream for the Treatment of Atopic Dermatitis
Brief Title: A Dose-Finding Study of GSK2894512 Cream in Subjects With Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203121
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-08

CONDITIONS: Dermatitis, Atopic
Keywords: Vehicle-Controlled; GSK2894512; Double blind; Dose-finding; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tapinarof

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- GSK2894512 1% cream twice daily (Experimental): Subjects will apply a thin layer of GSK2894512 1% (10 milligram per gram [mg/g]) topical cream twice daily (morning and evening) for 12 weeks, to all atopic dermatitis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 1% Cream
- GSK2894512 1% cream once daily (Experimental): Subjects will apply a thin layer of GSK2894512 1% (10 mg/g) topical cream once daily (evening) for 12 weeks, to all atopic dermatitis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 1% Cream
- GSK2894512 0.5% cream twice daily (Experimental): Subjects will apply a thin layer of GSK2894512 0.5% (5 mg/g) topical cream twice daily (morning and evening) for 12 weeks, to all atopic dermatitis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 0.5% Cream
- GSK2894512 0.5% cream once daily (Experimental): Subjects will apply a thin layer of GSK2894512 0.5% (5 mg/g) topical cream once daily (evening) for 12 weeks, to all atopic dermatitis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 0.5% Cream
- Vehicle cream twice daily (Placebo Comparator): Subjects will apply a thin layer of vehicle topical cream twice daily (morning and evening) for 12 weeks, to all atopic dermatitis lesions (except on the scalp).
  Interventions: Drug: Vehicle cream
- Vehicle cream once daily (Placebo Comparator): Subjects will apply a thin layer of vehicle topical cream once daily (evening) for 12 weeks, to all atopic dermatitis lesions (except on the scalp).
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: GSK2894512 1% Cream — 1.0% (10 mg/g) GSK2894512 will be supplied as white to off-white cream to be applied topically
  Arms: GSK2894512 1% cream once daily; GSK2894512 1% cream twice daily
Drug: GSK2894512 0.5% Cream — 0.5% (5 mg/g) GSK2894512 will be supplied as white to off-white cream to be applied topically
  Arms: GSK2894512 0.5% cream once daily; GSK2894512 0.5% cream twice daily
Drug: Vehicle cream — White to off-white vehicle cream base to be applied topically
  Arms: Vehicle cream once daily; Vehicle cream twice daily

SUMMARY:
This study will evaluate the efficacy and safety of two concentrations (0.5 percent [%] and 1%) and two application frequencies (once a day and twice a day) of GSK2894512 cream for the topical treatment in adolescent and adult subjects with atopic dermatitis. Results from this study will be considered when selecting the most appropriate concentration of GSK2894512 cream and application frequency in future clinical studies. This is a multicenter (United States, Canada, and Japan), randomized, double-blind (sponsor-unblind), vehicle-controlled, 6-arm, parallel-group, dose-finding study in adolescent and adult subjects with atopic dermatitis. Two concentrations of GSK2894512 cream (0.5% and 1%) and a vehicle control cream will be equally randomized and evaluated following application to all atopic dermatitis lesions (except on the scalp) once daily (evening) or twice daily (morning and evening) for 12 weeks. This study will consist of 3 periods: up to 4 weeks screening, 12 weeks double-blind treatment, and 4 weeks post-treatment follow-up. The total duration of subject participation will be approximately 16 to 20 weeks. Approximately 270 adolescent and adult males and females subjects with atopic dermatitis will be screened in order to have at least 228 randomized subjects (38 subjects for each of the 6 treatment groups) and approximately 204 evaluable subjects overall. Approximately 30 subjects will be randomized in Japan to achieve at least 24 evaluable Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 12 and 65 years of age inclusive, at the time of signing the informed consent
* Diagnosis of atopic dermatitis according to Hanifin and Rajka criteria and having active inflammation.
* Body surface area involvement >=5% and <=35%, excluding scalp, at Screening and Baseline.
* An IGA of atopic dermatitis score of >=3 at Baseline.
* At least one target lesion that measure at least 3 centimetre (cm) х 3 cm in size at Screening and Baseline and must be representative of the subject's disease state, but not located on the hands, feet, or genitalia.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: 1) Pre-menopausal females with one of the following procedures documented: tubal ligation; hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; bilateral oophorectomy. 2) Post-menopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone and estradiol levels consistent with menopause and falling into the central laboratory's postmenopausal reference range is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt are required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment; Reproductive potential and agrees to follow one of the options listed in the modified list of highly effective methods for avoiding pregnancy in females of reproductive potential from 30 days prior to the first dose of study medication and until after the last dose of study medication and completion of the follow-up visit.

Exclusion Criteria:

* Unstable course of atopic dermatitis (spontaneously improving or rapidly deteriorating) as determined by the investigator over the previous 4 weeks prior to Baseline.
* Concurrent conditions and history of other diseases: 1) Immunocompromized (eg, lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich Syndrome) or have a history of malignant disease within 5 years before the baseline visit; 2) Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks before the baseline visit; 3) Active acute bacterial, fungal, or viral (eg, herpes simplex, herpes zoster, chicken pox) skin infection within 1 week before the baseline visit; 4) Any other concomitant skin disorder (eg, generalized erythroderma such as Netherton's Syndrome, or psoriasis); pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of AD lesions or compromise subject safety; 5) Presence of AD lesions only on the hands or feet without prior history of involvement of other classical areas of involvement such as the face or the folds; 6) Other types of eczema.
* A history or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, may interfere with the subject's completion of the study.
* Known hypersensitivity to study treatment excipients.
* Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result within 3 months of screening.
* Liver function tests: alanine aminotransferase (ALT) >=2x upper limit of normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTc >=450 milliseconds (msec) or QTc >=480 msec for subjects with bundle branch block.

NOTES: The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF), with machine over-read. The QTc should be based on a single ECG obtained over a brief recording period. If QTc is outside of the threshold value, triplicate ECGs may be performed with the QTc values averaged.

* Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 4 weeks prior to the baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the subject's atopic dermatitis.
* Used any of the following treatments within the indicated washout period before the baseline visit: 12 weeks or 5 half-lives (whichever is longer) - biologic agents (eg, 18 weeks for omalizumab); 8 weeks - cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg, mycophenolate or tacrolimus); 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs; 2 weeks - topical treatments: corticosteroids, calcineurin inhibitors, or coal tar (on the body); 2 weeks - immunizations; sedating antihistamines (non sedating antihistamines are permitted); 1 week - topical antibiotics, antibacterial cleansing body wash/soap or diluted sodium hypochlorite "bleach" baths.
* Participated in a clinical study and received an investigational product within the following time period prior to the baseline visit: 4 weeks, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of alcohol or other substance abuse within the last 2 years.
* Participated in a previous study using GSK2894512 (or WBI-1001).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2015-12-01; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (33):
  - GSK Investigational Site, Fort Smith, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, North Logan, Connecticut
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, West Dundee, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Andover, Massachusetts
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, West Bloomfield, Michigan
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Saint Joseph, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Cranston, Rhode Island
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Seattle, Washington
- Canada (10):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Markham, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Richmond Hill, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Drummondville, Quebec
  - GSK Investigational Site, Québec, Quebec
- Japan (6):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants entered a 4 weeks screening phase and participants who met the eligibility criteria entered into the 12 weeks double-blind treatment phase and 4 weeks post-treatment follow-up phase. The total duration of participation in the study was 16 to 20 weeks.
Pre-assignment Details: A total of 363 adolescent and adult participants with atopic dermatitis (AD) were screened, of which 116 were screen failures and 247 entered the treatment phase. Participants in the treatment phase were randomized to receive GSK2894512 cream (0.5 or 1%) or vehicle control once daily (QD) or twice daily (BID).
Groups:
- GSK2894512 1% BID: Participants received 1% of GSK2894512 cream BID applied to all AD lesions via topical route for 12 weeks.
- GSK2894512 1% QD: Participants received 1% of GSK2894512 cream QD applied to all AD lesions via topical route for 12 weeks.
- GSK2894512 0.5% BID: Participants received 0.5% of GSK 2894512 cream BID applied to all AD lesions via topical route for 12 weeks.
- GSK2894512 0.5% QD: Participants received 0.5% of GSK2894512 cream QD applied to all AD lesions via topical route for 12 weeks.
- Vehicle BID: Participants received vehicle control cream BID applied to all AD lesions via topical route for 12 weeks.
- Vehicle QD: Participants received vehicle control cream QD applied to all AD lesions via topical route for 12 weeks.
Period: Overall Study
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Started | 40 | 41 | 43 | 41 | 42 | 40
Completed | 34 | 36 | 31 | 35 | 27 | 28
Not Completed | 6 | 5 | 12 | 6 | 15 | 12
Not completed — Adverse Event | 1 | 0 | 4 | 1 | 4 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Reached stopping criteria | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 4 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 3 | 3 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD | Total
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40 | 247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.5 (13.90) | 31.6 (15.72) | 29.0 (15.91) | 29.3 (14.02) | 27.9 (14.72) | 29.4 (15.15) | 29.3 (14.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 24 | 17 | 22 | 23 | 17 | 121
  Male | 22 | 17 | 26 | 19 | 19 | 23 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, Customized: White/Caucasian | 16 | 18 | 17 | 17 | 20 | 12 | 100
  Race/Ethnicity, Customized: Black/African American | 7 | 10 | 11 | 12 | 6 | 12 | 58
  Race/Ethnicity, Customized: American Indian/Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race/Ethnicity, Customized: Asian/S.E. Asian Descent/Japanese | 15 | 13 | 13 | 10 | 15 | 14 | 80
  Race/Ethnicity, Customized: American Indian/Alaska Native and African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race/Ethnicity, Customized: Asian/S.E. Asian/Japanese and African American | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Race/Ethnicity, Customized: Asian/S.E. Asian/Japanese and Black and White | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Race/Ethnicity, Customized: Asian/S.E. Asian/Japanese and White/Caucasian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Race/Ethnicity, Customized: Black/African American and White/Caucasian | 1 | 0 | 0 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have an Investigator Global Assessment (IGA) Score of Clear or Almost Clear (0 or 1) at Week 12 and a Minimum 2 Grade Improvement in IGA Score From Baseline to Week 12 for Intent to Treat (ITT) Population
Description: The IGA is a clinical tool for assessing the current state/severity of a participant's AD. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines. The percentage of participants who have an IGA score of clear or almost clear at Week 12 and a minimum 2 grade improvement from Baseline to Week 12 in IGA score was presented. . The analysis was performed on ITT Population which comprised of all randomized participants.
Time Frame: Baseline and up to Week 12
Population: ITT Population. Only those participants with data available at specified data points were analyzed.
Measure: Number; unit: Percentage of participant
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
Percentage of participant | 58 | 51 | 50 | 40 | 36 | 44
Statistical Analysis 1: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 22.6, 95% CI 2-sided [-2.4 to 45.5] — Difference between GSK2894512 1 percent BID and Vehicle BID has been presented
Statistical Analysis 2: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 7.4, 95% CI 2-sided [-18.3 to 32.0] — Difference between GSK2894512 1 percent QD and Vehicle QD has been presented
Statistical Analysis 3: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 14.3, 95% CI 2-sided [-11.2 to 38.7] — Difference between GSK2894512 0.5 percent BID and Vehicle BID has been presented
Statistical Analysis 4: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = -4.0, 95% CI 2-sided [-29.3 to 21.6] — Difference between GSK2894512 0.5 percent QD and Vehicle QD has been presented

2. Secondary Outcome: Mean Change From Baseline in Weekly Average of Daily Itch/Pruritus (Numeric Rating Scale [NRS]) Score
Description: NRS is a 11-point tool ranging from 0 (absent) to 10 (worst imaginable) to assess the severity of 11 disease-related signs and symptoms including itching, discoloration, bleeding, oozing, cracking, scaling, flaking, dry/rough, painful, burning, and stinging. Participants were asked to complete the self-administered sign and symptom severity diary containing NRS using a recall period of the past 24 hours. Question 1 of the diary was used to assess itch. Mean change from Baseline to Week 12 in weekly average of daily itch/pruritus based on the NRS was presented using mean and standard deviation (SD). Baseline was defined as the latest assessment prior to first dose and Change from Baseline was defined as post-dose weekly average value minus Baseline value.
Time Frame: Baseline and up to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Scores on a scale | -3.06 (2.657) | -3.10 (2.493) | -3.52 (2.307) | -3.39 (2.297) | -0.95 (2.107) | -3.50 (2.742)

3. Secondary Outcome: Mean Percent Change From Baseline in Weekly Average of Daily Itch/Pruritus NRS Score
Description: NRS is a 11-point tool ranging from 0 (absent) to 10 (worst imaginable) to assess the severity of 11 disease-related signs and symptoms including itching, discoloration, bleeding, oozing, cracking, scaling, flaking, dry/rough, painful, burning, and stinging. Participants were asked to complete the self-administered sign and symptom severity diary containing NRS using a recall period of the past 24 hours. Question 1 of the diary was used to assess itch. Mean percent change in weekly average of daily itch/pruritus based on the NRS was presented using mean and SD from Baseline to Week 12. Baseline was defined as the latest assessment prior to first dose and Change from Baseline was defined as post-dose weekly average value minus Baseline value.
Time Frame: Baseline and up to Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage Change | -64.69 (36.916) | -58.34 (45.632) | -60.39 (44.314) | -61.40 (34.958) | -29.16 (55.251) | -55.62 (40.320)

4. Secondary Outcome: Percentage of Participants Who Achieve a Minimum 3- Point Improvement in Itch/Pruritus (NRS) From Baseline to Each Study Visit
Description: NRS is a 11-point tool ranging from 0 (absent) to 10 (worst imaginable) to assess the severity of 11 disease-related signs and symptoms including itching, discoloration, bleeding, oozing, cracking, scaling, flaking, dry/rough, painful, burning, and stinging. Participants were asked to complete the self-administered sign and symptom severity diary containing NRS using a recall period of the past 24 hours. Question 1 of the diary was used to assess itch. Percentage of participants who achieved a minimum 3-point improvement in itch/pruritus (NRS) from Baseline to each study visit were measured. Baseline was defined as the latest assessment prior to first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Week 1, 2, 4, 8, 12, 14, 16, early withdrawal (EW) (up to Week 16)
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage of Participants
  Week 1; n= 29,35,33,31,24,25: number analyzed (Participants) | 29 | 35 | 33 | 31 | 24 | 25
  Week 1; n= 29,35,33,31,24,25 | 24 | 9 | 9 | 16 | 8 | 12
  Week 2; n= 28,30,36,30,26,23: number analyzed (Participants) | 28 | 30 | 36 | 30 | 26 | 23
  Week 2; n= 28,30,36,30,26,23 | 36 | 33 | 22 | 33 | 12 | 22
  Week 4; n= 31,31,29,31,20,25: number analyzed (Participants) | 31 | 31 | 29 | 31 | 20 | 25
  Week 4; n= 31,31,29,31,20,25 | 42 | 48 | 45 | 52 | 35 | 28
  Week 8; n= 26,26,29,30,21,23: number analyzed (Participants) | 26 | 26 | 29 | 30 | 21 | 23
  Week 8; n= 26,26,29,30,21,23 | 46 | 50 | 48 | 57 | 29 | 30
  Week 12; n= 22,25,23,23,14,16: number analyzed (Participants) | 22 | 25 | 23 | 23 | 14 | 16
  Week 12; n= 22,25,23,23,14,16 | 55 | 52 | 61 | 52 | 14 | 38
  Week 14; n= 21,20,19,20,17,14: number analyzed (Participants) | 21 | 20 | 19 | 20 | 17 | 14
  Week 14; n= 21,20,19,20,17,14 | 38 | 40 | 58 | 50 | 29 | 50
  Week 16; n= 15,14,22,17,12,13: number analyzed (Participants) | 15 | 14 | 22 | 17 | 12 | 13
  Week 16; n= 15,14,22,17,12,13 | 33 | 21 | 41 | 47 | 17 | 23
  EW; n= 0,3,2,2,5,6: number analyzed (Participants) | 0 | 3 | 2 | 2 | 5 | 6
  EW; n= 0,3,2,2,5,6 |  | 0 | 50 | 50 | 0 | 17

5. Secondary Outcome: Mean Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: The EASI scoring system is a standard clinical tool for assessing the severity of AD that takes into account the overall severity of erythema, infiltration/papulation, excoriation, and lichenification, as well as the extent of BSA affected with AD. These 4 clinical signs were graded on a 4-point scale (0 [absent] to 3 [severe]) for each of the 4 specified body regions (head and neck, upper extremities, lower extremities, and trunk). Body area involvement ranged from 0 (0%) to 6 (90-100%). Total EASI score was calculated as a sum of scores of all 4 specified body region. Range for EASI total score is 0 (absent) to 72 (severe). Baseline was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. Mean change from Baseline was presented in the form of mean and SD. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Week 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Scores on a scale
  Week 1; n= 38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38,41,39,37,38,32 | -2.58 (3.965) | -3.83 (4.410) | -3.22 (3.585) | -2.51 (3.240) | -1.84 (2.730) | -1.06 (3.660)
  Week 2; n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39,39,39,39,33,32 | -4.89 (4.052) | -5.69 (3.996) | -5.27 (3.848) | -4.21 (3.337) | -3.18 (3.545) | -1.67 (3.079)
  Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38,39,38,39,30,32 | -6.55 (3.808) | -7.18 (4.534) | -7.42 (3.749) | -6.19 (3.588) | -4.45 (4.180) | -2.94 (3.788)
  Week 8; n= 36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36,37,34,38,29,27 | -7.00 (4.759) | -8.12 (4.924) | -8.67 (5.039) | -7.62 (4.539) | -5.24 (5.267) | -4.15 (5.190)
  Week 12; n= 36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36,37,32,35,28,25 | -7.85 (5.000) | -8.16 (4.931) | -10.12 (4.665) | -8.16 (5.077) | -6.05 (5.937) | -5.58 (5.668)
  Week 14; n= 34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34,35,31,33,27,25 | -7.08 (3.955) | -7.36 (4.683) | -9.07 (5.367) | -7.42 (4.798) | -6.28 (5.335) | -5.44 (5.050)
  Week 16; n= 34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34,36,31,35,27,25 | -6.45 (4.245) | -7.45 (5.106) | -8.85 (5.654) | -7.67 (4.405) | -6.29 (6.158) | -5.40 (5.315)
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | -1.03 (5.523) | 3.40 (4.023) | 3.11 (9.042) | -2.97 (6.661) | 2.01 (4.418) | 3.38 (9.746)

6. Secondary Outcome: Mean Percent Change From Baseline in EASI Score
Description: The EASI scoring system is a standard clinical tool for assessing the severity of AD that takes into account the overall severity of erythema, infiltration/papulation, excoriation, and lichenification, as well as the extent of BSA affected with AD. These 4 clinical signs were graded on a 4-point scale (0 [absent] to 3 [severe]) for each of the 4 specified body regions (head and neck, upper extremities, lower extremities, and trunk). Body area involvement ranged from 0 (0%) to 6 (90-100%). Total EASI score was calculated as a sum of scores of all 4 specified body region. Range for EASI total score is 0 (absent) to 72 (severe). Baseline was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. Mean percent change from Baseline was presented in the form of mean and SD. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage Change
  Week 1; n= 38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38,41,39,37,38,32 | -23.83 (42.885) | -34.76 (32.718) | -24.19 (21.716) | -25.81 (28.724) | -16.79 (25.777) | -7.51 (36.549)
  Week 2; n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39,39,39,39,33,32 | -48.70 (33.089) | -54.21 (29.107) | -42.60 (26.428) | -40.41 (30.835) | -32.03 (32.737) | -13.98 (38.616)
  Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38,39,38,39,30,32 | -64.95 (23.948) | -66.40 (30.182) | -60.07 (23.967) | -55.38 (24.465) | -40.74 (30.097) | -30.54 (36.196)
  Week 8; n= 36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36,37,34,38,29,27 | -68.14 (28.052) | -73.57 (27.204) | -70.52 (25.062) | -65.12 (26.089) | -50.78 (33.026) | -43.15 (41.388)
  Week 12; n= 36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36,37,32,35,28,25 | -77.19 (28.152) | -73.02 (25.068) | -80.13 (18.602) | -69.49 (24.805) | -56.73 (38.234) | -60.29 (34.253)
  Week 14; n= 34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34,35,31,33,27,25 | -71.15 (27.875) | -65.53 (29.777) | -70.37 (31.907) | -64.72 (25.594) | -60.26 (31.632) | -55.21 (31.514)
  Week 16; n= 34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34,36,31,35,27,25 | -63.59 (36.461) | -63.70 (25.833) | -69.89 (32.687) | -67.28 (25.745) | -57.52 (47.140) | -52.47 (38.236)
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | -0.83 (98.753) | 42.27 (43.950) | 8.74 (87.714) | -35.40 (66.349) | 13.69 (32.424) | 32.55 (86.387)

7. Secondary Outcome: Percentage of Participants With a Minimum 2-grade Improvement in IGA Score From Baseline to Each Visit
Description: The IGA is a clinical tool for assessing the current state/severity of a participant's AD. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines. IGA is made without reference to previous scores. The percentage of participants with a minimum 2-grade improvement in IGA score from Baseline at Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and early withdrawal (EW) visit was presented in the form of mean and SD. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage of participants
  Week 1; n= 38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38,41,39,37,38,32 | 5 | 7 | 0 | 3 | 5 | 6
  Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39, 39, 39, 39, 33, 32 | 18 | 21 | 10 | 15 | 15 | 9
  Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38,39,38,39,30,32 | 32 | 46 | 26 | 28 | 23 | 13
  Week 8; n= 36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36,37,34,38,29,27 | 44 | 59 | 38 | 45 | 28 | 22
  Week 12; n= 36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36,37,32,35,28,25 | 64 | 51 | 53 | 43 | 39 | 44
  Week 14; n= 34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34,35,31,33,27,25 | 47 | 46 | 55 | 42 | 26 | 36
  Week 16; n= 34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34,36,31,35,27,25 | 35 | 36 | 39 | 43 | 33 | 32
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | 33 | 0 | 14 | 33 | 0 | 9

8. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 at Each Visit
Description: The IGA is a clinical tool for assessing the current state/severity of a participant's AD. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines. IGA is made without reference to previous scores. The percentage of participants with an IGA score of 0 or 1 at Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and EW visit was presented in the form of mean and SD. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage of participants
  Week 1; 38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; 38,41,39,37,38,32 | 5 | 5 | 0 | 3 | 3 | 3
  Week 2; n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39,39,39,39,33,32 | 18 | 18 | 10 | 13 | 15 | 9
  Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38,39,38,39,30,32 | 32 | 38 | 26 | 23 | 20 | 9
  Week 8; n= 36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36,37,34,38,29,27 | 42 | 54 | 38 | 42 | 28 | 19
  Week 12; n= 36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36,37,32,35,28,25 | 58 | 51 | 50 | 40 | 36 | 44
  Week 14; n= 34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34,35,31,33,27,25 | 44 | 43 | 52 | 36 | 26 | 36
  Week 16; n= 34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34,36,31,35,27,25 | 35 | 36 | 39 | 40 | 30 | 28
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | 33 | 0 | 14 | 33 | 0 | 9

9. Secondary Outcome: Percentage of Participants With >=50 Percent Improvement From Baseline in EASI
Description: The EASI scoring system is a standard clinical tool for assessing the severity of AD that takes into account the overall severity of erythema, infiltration/papulation, excoriation, and lichenification, as well as the extent of BSA affected with AD. These 4 clinical signs were graded on a 4-point scale for each of the 4 specified body regions (head and neck, upper extremities, lower extremities, and trunk). Percentage of participants with >=50 percent improvement in EASI score from Baseline to Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and EW were presented and statistical analysis was performed using a repeated measures factorial logistic regression model. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage of participants
  Week 1; n= 38, 41, 39, 37, 38, 32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38, 41, 39, 37, 38, 32 | 32 | 39 | 13 | 22 | 11 | 13
  Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39, 39, 39, 39, 33, 32 | 56 | 56 | 38 | 36 | 33 | 19
  Week 4; n= 38, 39, 38, 39, 30, 32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38, 39, 38, 39, 30, 32 | 76 | 72 | 63 | 59 | 37 | 41
  Week 8; n= 36, 37, 34, 38, 29, 27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36, 37, 34, 38, 29, 27 | 81 | 92 | 85 | 79 | 59 | 56
  Week 12; n= 36, 37, 32, 35, 28, 25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36, 37, 32, 35, 28, 25 | 83 | 84 | 97 | 74 | 64 | 84
  Week 14; n= 34, 35, 31, 33, 27, 25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34, 35, 31, 33, 27, 25 | 85 | 74 | 81 | 76 | 63 | 68
  Week 16; n= 34, 36, 31 35, 27, 25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34, 36, 31 35, 27, 25 | 76 | 78 | 84 | 71 | 67 | 72
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | 33 | 0 | 29 | 33 | 0 | 9
Statistical Analysis 1: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 21.1, 95% CI 2-sided [-2.7 to 43.1] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 1 has been presented
Statistical Analysis 2: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 26.5, 95% CI 2-sided [3.3 to 47.5] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 1 has been presented
Statistical Analysis 3: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 2.3, 95% CI 2-sided [-19.5 to 24.5] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 1 has been presented
Statistical Analysis 4: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 9.1, 95% CI 2-sided [-14.5 to 32.0] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 1 has been presented
Statistical Analysis 5: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 23.1, 95% CI 2-sided [-0.3 to 44.6] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 6: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 37.7, 95% CI 2-sided [14.7 to 57.6] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 7: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 5.1, 95% CI 2-sided [-18.0 to 27.8] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 8: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 17.1, 95% CI 2-sided [-6.4 to 39.0] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 9: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 39.6, 95% CI 2-sided [16.0 to 60.0] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 10: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 31.2, 95% CI 2-sided [7.8 to 52.1] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 11: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 26.5, 95% CI 2-sided [2.3 to 48.4] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 12: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 18.3, 95% CI 2-sided [-5.3 to 40.5] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 13: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 21.9, 95% CI 2-sided [-2.3 to 44.7] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 14: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 36.3, 95% CI 2-sided [12.1 to 57.6] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 15: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 26.7, 95% CI 2-sided [1.7 to 49.0] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 16: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 23.4, 95% CI 2-sided [-1.5 to 46.1] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 17: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 19.0, 95% CI 2-sided [-6.0 to 42.3] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 18: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = -0.2, 95% CI 2-sided [-25.0 to 25.0] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 19: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 32.6, 95% CI 2-sided [6.9 to 55.0] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 20: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = -9.7, 95% CI 2-sided [-34.6 to 16.1] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 21: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 22.3, 95% CI 2-sided [-3.1 to 45.3] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 22: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 6.3, 95% CI 2-sided [-19.5 to 31.5] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 23: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 17.7, 95% CI 2-sided [-8.4 to 41.9] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 24: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 7.8, 95% CI 2-sided [-17.8 to 33.1] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 25: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 9.8, 95% CI 2-sided [-15.5 to 33.9] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 26: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 5.8, 95% CI 2-sided [-19.7 to 30.5] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 27: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 17.2, 95% CI 2-sided [-9.0 to 41.4] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 28: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = -0.6, 95% CI 2-sided [-26.0 to 25.0] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 29: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 33.3, 95% CI 2-sided [-31.9 to 90.6] — Difference between GSK2894512 1 % BID and Vehicle BID at EW has been presented
Statistical Analysis 30: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = -9.1, 95% CI 2-sided [-62.4 to 47.8] — Difference between GSK2894512 1 % QD and Vehicle QD at EW has been presented
Statistical Analysis 31: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 28.6, 95% CI 2-sided [-19.2 to 71.0] — Difference between GSK2894512 0.5 % BID and Vehicle BID at EW has been presented
Statistical Analysis 32: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 24.2, 95% CI 2-sided [-40.3 to 80.9] — Difference between GSK2894512 0.5 % QD and Vehicle QD at EW has been presented

10. Secondary Outcome: Percentage of Participants With >=75 Percent Improvement From Baseline in EASI
Description: The EASI scoring system is a standard clinical tool for assessing the severity of AD that takes into account the overall severity of erythema, infiltration/papulation, excoriation, and lichenification, as well as the extent of BSA affected with AD. These 4 clinical signs were graded on a 4-point scale for each of the 4 specified body regions (head and neck, upper extremities, lower extremities, and trunk). Percentage of participants with >=75 percent improvement in EASI score from Baseline to Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and EW were presented and statistical analysis was performed using a repeated measures factorial logistic regression model. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage of participants
  Week 1; n= 38, 41, 39, 37, 38, 32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38, 41, 39, 37, 38, 32 | 5 | 12 | 0 | 5 | 0 | 6
  Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39, 39, 39, 39, 33, 32 | 21 | 33 | 13 | 21 | 9 | 3
  Week 4; n= 38, 39, 38, 39, 30, 32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38, 39, 38, 39, 30, 32 | 37 | 51 | 29 | 26 | 20 | 9
  Week 8; n= 36, 37, 34, 38, 29, 27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36, 37, 34, 38, 29, 27 | 44 | 57 | 53 | 37 | 31 | 26
  Week 12; n= 36, 37, 32, 35, 28, 25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36, 37, 32, 35, 28, 25 | 67 | 57 | 69 | 46 | 39 | 40
  Week 14; n= 34, 35, 31, 33, 27, 25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34, 35, 31, 33, 27, 25 | 50 | 49 | 68 | 36 | 41 | 36
  Week 16; n= 34, 36, 31 35, 27, 25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34, 36, 31 35, 27, 25 | 47 | 39 | 61 | 43 | 44 | 32
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | 33 | 0 | 14 | 33 | 0 | 9
Statistical Analysis 1: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 5.3, 95% CI 2-sided [-18.3 to 28.4] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 1 has been presented
Statistical Analysis 2: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 5.9, 95% CI 2-sided [-17.1 to 28.4] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 1 has been presented
Statistical Analysis 3: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = -0.8, 95% CI 2-sided [-24.0 to 22.7] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 1 has been presented
Statistical Analysis 4: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 11.4, 95% CI 2-sided [-12.0 to 33.9] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 5: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 30.2, 95% CI 2-sided [6.8 to 51.0] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 6: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 3.7, 95% CI 2-sided [-19.4 to 26.6] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 7: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 17.4, 95% CI 2-sided [-6.0 to 39.5] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 8: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 16.8, 95% CI 2-sided [-7.1 to 39.4] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 9: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 41.9, 95% CI 2-sided [19.2 to 61.2] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 10: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 8.9, 95% CI 2-sided [-14.9 to 32.0] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 11: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 16.3, 95% CI 2-sided [-7.3 to 38.3] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 12: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 13.4, 95% CI 2-sided [-11.3 to 36.5] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 13: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 30.8, 95% CI 2-sided [6.1 to 52.8] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 14: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 21.9, 95% CI 2-sided [-3.0 to 44.9] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 15: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 10.9, 95% CI 2-sided [-13.5 to 34.7] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 16: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 27.4, 95% CI 2-sided [2.5 to 49.9] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 17: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 16.8, 95% CI 2-sided [-9.0 to 40.7] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 18: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 29.5, 95% CI 2-sided [3.7 to 52.3] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 19: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 5.7, 95% CI 2-sided [-20.1 to 30.9] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 20: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 9.3, 95% CI 2-sided [-16.2 to 33.8] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 21: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 12.6, 95% CI 2-sided [-13.4 to 37.3] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 22: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 27.0, 95% CI 2-sided [0.7 to 50.5] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 23: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 0.4, 95% CI 2-sided [-25.6 to 25.6] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 24: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 2.6, 95% CI 2-sided [-22.6 to 27.6] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 25: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 6.9, 95% CI 2-sided [-18.7 to 31.7] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 26: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 16.8, 95% CI 2-sided [-9.5 to 41.4] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 27: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 10.9, 95% CI 2-sided [-14.9 to 35.8] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 28: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 33.3, 95% CI 2-sided [-31.9 to 90.6] — Difference between GSK2894512 1 % BID and Vehicle BID at EW has been presented
Statistical Analysis 29: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = -9.1, 95% CI 2-sided [-62.4 to 47.8] — Difference between GSK2894512 1 % QD and Vehicle QD at EW has been presented
Statistical Analysis 30: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = 14.3, 95% CI 2-sided [-32.2 to 57.9] — Difference between GSK2894512 0.5 % BID and Vehicle BID at EW has been presented
Statistical Analysis 31: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 24.2, 95% CI 2-sided [-40.3 to 80.9] — Difference between GSK2894512 0.5 % QD and Vehicle QD at EW has been presented

11. Secondary Outcome: Mean Change From Baseline in Total Severity Score (TSS)
Description: A target lesion of at least 3 centimeter square (cm^2) was selected at Baseline. The severity of the following signs: erythema, induration/papulation, lichenification, oozing/crusting, and scaling was assessed on a 4-point scale ranging from 0 (absent) to 3 (severe), with higher values indicating greater severity of symptoms. TSS (maximum score 15) was calculated based on these signs. Mean change from Baseline in TSS at Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and EW visit was presented using mean and SD. Baseline value was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Scores on a scale
  Week 1; n= 38, 41, 39, 37, 38, 32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38, 41, 39, 37, 38, 32 | -1.8 (2.04) | -2.7 (2.75) | -2.1 (1.81) | -1.8 (2.02) | -1.9 (2.60) | -0.9 (2.21)
  Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39, 39, 39, 39, 33, 32 | -3.6 (2.50) | -4.0 (2.42) | -3.7 (2.45) | -3.3 (2.46) | -3.1 (2.73) | -1.8 (2.73)
  Week 4; n= 38, 39, 38, 39, 30, 32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38, 39, 38, 39, 30, 32 | -4.2 (2.48) | -4.5 (2.39) | -5.1 (2.58) | -4.1 (2.64) | -3.3 (2.68) | -3.0 (3.03)
  Week 8; n= 36, 37, 34, 38, 29, 27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36, 37, 34, 38, 29, 27 | -4.7 (2.37) | -5.4 (2.65) | -6.1 (2.17) | -5.1 (2.34) | -4.7 (2.68) | -4.3 (3.01)
  Week 12; n= 36, 37, 32, 35, 28, 25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36, 37, 32, 35, 28, 25 | -5.8 (2.92) | -5.5 (2.64) | -7.0 (2.38) | -5.5 (2.58) | -4.6 (2.64) | -5.2 (2.97)
  Week 14; n= 34, 35, 31, 33, 27, 25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34, 35, 31, 33, 27, 25 | -5.6 (2.67) | -5.1 (2.19) | -5.5 (3.22) | -4.4 (3.09) | -5.0 (2.72) | -5.0 (2.88)
  Week 16; n= 34, 36, 31, 35, 27, 25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34, 36, 31, 35, 27, 25 | -5.4 (2.98) | -4.9 (2.27) | -6.0 (2.91) | -5.1 (2.65) | -4.8 (2.62) | -4.9 (2.74)
  EW; n= 3, 4, 7, 3, 11, 11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3, 4, 7, 3, 11, 11 | -2.3 (4.93) | 0.5 (5.26) | -0.4 (4.83) | -2.7 (3.51) | -1.1 (3.65) | -0.1 (4.04)

12. Secondary Outcome: Mean Percent Change From Baseline in TSS
Description: A target lesion of at least 3 cm^2 was selected at Baseline. The severity of the following signs: erythema, induration/papulation, lichenification, oozing/crusting, and scaling was assessed on a 4-point scale ranging from 0 (absent) to 3 (severe) , with higher values indicating greater severity of symptoms. TSS (maximum score 15) was calculated based on these signs. Mean percent change from Baseline in TSS at Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and EW visit was presented using mean and SD. Baseline value was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Week 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage Change
  Week 1; n= 38, 41, 39, 37, 38, 32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38, 41, 39, 37, 38, 32 | -23.5 (27.99) | -33.7 (31.01) | -25.8 (21.94) | -22.6 (24.78) | -22.0 (27.47) | -9.8 (28.06)
  Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39, 39, 39, 39, 33, 32 | -46.7 (32.75) | -52.8 (28.45) | -44.5 (26.15) | -42.4 (33.54) | -35.1 (29.29) | -17.6 (40.06)
  Week 4; n= 38, 39, 38, 39, 30, 32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38, 39, 38, 39, 30, 32 | -55.8 (31.18) | -60.1 (28.58) | -60.3 (27.68) | -52.1 (33.85) | -37.4 (27.29) | -33.5 (36.16)
  Week 8; n= 36, 37, 34, 38, 29, 27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36, 37, 34, 38, 29, 27 | -61.7 (28.14) | -69.1 (27.56) | -71.0 (20.75) | -65.3 (28.31) | -57.4 (31.55) | -50.0 (35.53)
  Week 12; n= 36, 37, 32, 35, 28, 25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36, 37, 32, 35, 28, 25 | -74.3 (31.61) | -73.1 (31.69) | -80.9 (18.59) | -68.6 (27.17) | -56.2 (30.53) | -62.6 (30.39)
  Week 14; n= 34, 35, 31, 33, 27, 25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34, 35, 31, 33, 27, 25 | -73.5 (30.31) | -71.1 (29.53) | -63.0 (32.96) | -53.7 (35.25) | -59.7 (34.87) | -60.2 (29.97)
  Week 16; n= 34, 36, 31, 35, 27, 25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34, 36, 31, 35, 27, 25 | -69.3 (33.20) | -66.0 (30.03) | -68.8 (30.66) | -63.5 (29.78) | -59.8 (33.68) | -60.3 (31.16)
  EW; n= 3, 4, 7, 3, 11, 11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3, 4, 7, 3, 11, 11 | -26.7 (64.29) | 1.4 (82.20) | -2.9 (75.44) | -40.3 (56.57) | -7.9 (41.91) | 5.0 (59.63)

13. Secondary Outcome: Mean Change From Baseline in Individual Signs of TSS
Description: The severity of the following signs: erythema, induration/papulation, lichenification, oozing/crusting, and scaling was assessed on a 4-point scale ranging from 0 (absent) to 3 (severe) and TSS (maximum score 15) was calculated based on these signs. Mean change from Baseline in individual signs of TSS was presented using mean and SD. Baseline value was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. If the participant had more than 3 missing days during the week, then the weekly average was not calculated and treated as missing data and excluded from the analysis. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Scores on a scale
  Erythema; Week 1; n= 38, 41, 39, 37, 38, 32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Erythema; Week 1; n= 38, 41, 39, 37, 38, 32 | -0.6 (0.55) | -0.8 (0.88) | -0.4 (0.63) | -0.4 (0.55) | -0.4 (0.76) | -0.2 (0.66)
  Erythema; Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Erythema; Week 2; n= 39, 39, 39, 39, 33, 32 | -1.1 (0.70) | -1.1 (0.84) | -0.8 (0.76) | -0.7 (0.75) | -0.6 (0.78) | -0.3 (0.93)
  Erythema; Week 4; n= 38, 39, 38, 39, 30, 32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Erythema; Week 4; n= 38, 39, 38, 39, 30, 32 | -1.1 (0.69) | -1.3 (0.75) | -1.2 (0.79) | -0.9 (0.79) | -0.8 (0.73) | -0.6 (0.87)
  Erythema; Week 8; n= 36, 37, 34, 38, 29, 27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Erythema; Week 8; n= 36, 37, 34, 38, 29, 27 | -1.3 (0.70) | -1.5 (0.77) | -1.4 (0.61) | -1.2 (0.73) | -1.2 (0.85) | -0.9 (1.01)
  Erythema; Week 12; n= 36, 37, 32, 35, 28, 25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Erythema; Week 12; n= 36, 37, 32, 35, 28, 25 | -1.5 (0.84) | -1.5 (0.80) | -1.7 (0.69) | -1.3 (0.84) | -1.1 (0.77) | -1.0 (0.89)
  Erythema; Week 14; n= 34, 35, 31, 33, 27, 25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Erythema; Week 14; n= 34, 35, 31, 33, 27, 25 | -1.5 (0.83) | -1.4 (0.77) | -1.3 (0.97) | -1.0 (0.75) | -1.2 (0.74) | -1.0 (0.79)
  Erythema; Week 16; n= 34, 36 , 31, 35, 27, 25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Erythema; Week 16; n= 34, 36 , 31, 35, 27, 25 | -1.5 (0.83) | -1.3 (0.82) | -1.4 (0.92) | -1.1 (0.77) | -1.1 (0.87) | -1.0 (0.68)
  Erythema; EW; n= 3, 4, 7, 3, 11, 11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  Erythema; EW; n= 3, 4, 7, 3, 11, 11 | -0.7 (1.15) | -0.3 (0.96) | -0.4 (0.98) | -1.0 (1.00) | -0.4 (1.12) | -0.1 (1.38)
  Induration/Papulation;Week 1; n=38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Induration/Papulation;Week 1; n=38,41,39,37,38,32 | -0.3 (0.48) | -0.6 (0.77) | -0.5 (0.68) | -0.4 (0.60) | -0.3 (0.65) | -0.1 (0.55)
  Induration/Papulation;Week 2;n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Induration/Papulation;Week 2;n= 39,39,39,39,33,32 | -0.8 (0.73) | -1.0 (0.87) | -0.8 (0.84) | -0.8 (0.73) | -0.6 (0.87) | -0.4 (0.87)
  Induration/Papulation;Week 4;n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Induration/Papulation;Week 4;n= 38,39,38,39,30,32 | -1.0 (0.82) | -1.2 (0.86) | -1.1 (0.78) | -0.9 (0.83) | -0.7 (0.75) | -0.7 (0.79)
  Induration/Papulation;Week 8;n= 36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Induration/Papulation;Week 8;n= 36,37,34,38,29,27 | -1.1 (0.65) | -1.2 (1.00) | -1.4 (0.66) | -1.2 (0.69) | -1.0 (0.76) | -0.9 (0.75)
  Induration/Papulation;Week 12;n=36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Induration/Papulation;Week 12;n=36,37,32,35,28,25 | -1.4 (0.87) | -1.4 (0.86) | -1.6 (0.72) | -1.2 (0.73) | -0.8 (0.79) | -1.1 (0.86)
  Induration/Papulation;Week 14;n=34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Induration/Papulation;Week 14;n=34,35,31,33,27,25 | -1.3 (0.86) | -1.3 (0.64) | -1.3 (0.73) | -0.9 (0.83) | -0.9 (0.75) | -1.1 (0.83)
  Induration/Papulation;Week 16;n=34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Induration/Papulation;Week 16;n=34,36,31,35,27,25 | -1.2 (0.82) | -1.2 (0.74) | -1.4 (0.75) | -1.2 (0.82) | -0.8 (0.68) | -1.1 (0.91)
  Induration/Papulation; EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  Induration/Papulation; EW; n= 3,4,7,3,11,11 | -0.3 (1.53) | 0.0 (0.82) | -0.1 (1.35) | 0.0 (1.00) | -0.3 (1.19) | 0.1 (1.38)
  Lichenification; Week 1;n=38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Lichenification; Week 1;n=38,41,39,37,38,32 | -0.3 (0.63) | -0.5 (0.81) | -0.4 (0.60) | -0.4 (0.54) | -0.4 (0.63) | -0.2 (0.42)
  Lichenification; Week 2;n=39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Lichenification; Week 2;n=39,39,39,39,33,32 | -0.6 (0.81) | -0.8 (0.78) | -0.7 (0.66) | -0.7 (0.73) | -0.7 (0.78) | -0.4 (0.76)
  Lichenification; Week 4;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Lichenification; Week 4;n=38,39,38,39,30,32 | -0.8 (0.81) | -0.9 (0.70) | -1.1 (0.73) | -0.9 (0.84) | -0.6 (0.89) | -0.6 (0.88)
  Lichenification; Week 8;n=36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Lichenification; Week 8;n=36,37,34,38,29,27 | -0.9 (0.83) | -1.1 (0.80) | -1.2 (0.67) | -1.1 (0.74) | -0.9 (0.65) | -1.0 (0.76)
  Lichenification; Week 12;n=36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Lichenification; Week 12;n=36,37,32,35,28,25 | -1.2 (0.91) | -1.1 (0.75) | -1.5 (0.57) | -1.2 (0.75) | -1.0 (0.67) | -1.3 (0.74)
  Lichenification; Week 14;n=34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Lichenification; Week 14;n=34,35,31,33,27,25 | -1.2 (0.84) | -1.0 (0.71) | -1.2 (0.83) | -1.1 (0.70) | -1.0 (0.85) | -1.2 (0.82)
  Lichenification; Week 16;n=34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Lichenification; Week 16;n=34,36,31,35,27,25 | -1.1 (0.98) | -1.0 (0.70) | -1.3 (0.73) | -1.1 (0.72) | -1.0 (0.76) | -1.2 (0.65)
  Lichenification; EW;n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  Lichenification; EW;n= 3,4,7,3,11,11 | -0.7 (1.15) | 0.0 (0.82) | -0.4 (0.98) | -1.0 (1.00) | -0.4 (0.81) | -0.2 (0.98)
  Oozing/crusting; Week 1;n=38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Oozing/crusting; Week 1;n=38,41,39,37,38,32 | -0.2 (0.47) | -0.4 (0.62) | -0.4 (0.63) | -0.3 (0.47) | -0.3 (0.91) | -0.2 (0.68)
  Oozing/crusting; Week 2;n=39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Oozing/crusting; Week 2;n=39,39,39,39,33,32 | -0.5 (0.60) | -0.4 (0.55) | -0.7 (0.79) | -0.4 (0.55) | -0.5 (0.75) | -0.4 (0.66)
  Oozing/crusting; Week 4;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Oozing/crusting; Week 4;n=38,39,38,39,30,32 | -0.6 (0.65) | -0.5 (0.64) | -0.8 (0.86) | -0.6 (0.67) | -0.6 (0.82) | -0.5 (0.80)
  Oozing/crusting; Week 8;n=36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Oozing/crusting; Week 8;n=36,37,34,38,29,27 | -0.6 (0.64) | -0.6 (0.75) | -1.0 (0.90) | -0.7 (0.65) | -0.6 (0.78) | -0.7 (0.82)
  Oozing/crusting; Week 12;n=36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Oozing/crusting; Week 12;n=36,37,32,35,28,25 | -0.6 (0.60) | -0.6 (0.72) | -1.1 (0.93) | -0.7 (0.66) | -0.7 (0.81) | -0.8 (0.94)
  Oozing/crusting; Week 14;n=34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Oozing/crusting; Week 14;n=34,35,31,33,27,25 | -0.6 (0.65) | -0.5 (0.78) | -0.8 (1.00) | -0.5 (0.94) | -0.8 (0.79) | -0.9 (0.83)
  Oozing/crusting; Week 16;n=34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Oozing/crusting; Week 16;n=34,36,31,35,27,25 | -0.6 (0.61) | -0.6 (0.77) | -1.0 (1.03) | -0.7 (0.62) | -0.8 (0.75) | -0.8 (0.87)
  Oozing/crusting; EW;n=3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  Oozing/crusting; EW;n=3,4,7,3,11,11 | -0.3 (0.58) | 0.8 (1.50) | 0.6 (1.40) | 0.0 (0.00) | 0.0 (0.77) | 0.1 (0.70)
  Scaling; Week 1;n=38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Scaling; Week 1;n=38,41,39,37,38,32 | -0.3 (0.85) | -0.4 (0.70) | -0.4 (0.68) | -0.3 (0.78) | -0.4 (0.72) | -0.2 (0.63)
  Scaling; Week 2;n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Scaling; Week 2;n= 39,39,39,39,33,32 | -0.6 (0.82) | -0.7 (0.68) | -0.6 (0.67) | -0.6 (0.71) | -0.6 (0.78) | -0.3 (0.63)
  Scaling; Week 4;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Scaling; Week 4;n=38,39,38,39,30,32 | -0.8 (0.78) | -0.7 (0.69) | -0.8 (0.75) | -0.8 (0.81) | -0.7 (0.71) | -0.6 (0.87)
  Scaling; Week 8;n=36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Scaling; Week 8;n=36,37,34,38,29,27 | -0.8 (0.79) | -0.9 (0.66) | -1.1 (0.71) | -0.9 (0.71) | -1.0 (0.76) | -0.8 (0.88)
  Scaling; Week 12;n=36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Scaling; Week 12;n=36,37,32,35,28,25 | -1.1 (0.83) | -0.9 (0.70) | -1.2 (0.72) | -1.0 (0.80) | -1.0 (0.67) | -0.9 (0.91)
  Scaling; Week 14;n=34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Scaling; Week 14;n=34,35,31,33,27,25 | -1.0 (0.85) | -0.9 (0.73) | -1.0 (0.80) | -0.8 (0.87) | -1.0 (0.81) | -0.9 (0.88)
  Scaling; Week 16;n=34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Scaling; Week 16;n=34,36,31,35,27,25 | -1.0 (0.90) | -0.8 (0.75) | -1.0 (0.68) | -0.9 (0.74) | -1.1 (0.70) | -0.8 (0.80)
  Scaling; EW;n=3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  Scaling; EW;n=3,4,7,3,11,11 | -0.3 (0.58) | 0.0 (1.41) | 0.0 (0.82) | -0.7 (0.58) | -0.1 (1.04) | 0.0 (0.89)

14. Secondary Outcome: Mean Percent Change From Baseline in Individual Signs of TSS
Description: The severity of the following signs: erythema, induration/papulation, lichenification, oozing/crusting, and scaling was assessed on a 4-point scale ranging from 0 (absent) to 3 (severe) and TSS (maximum score 15) was calculated based on these signs. Mean percent change from Baseline in individual signs of TSS was presented using mean and SD. Baseline value was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. NA indicates that data were not available. If the participant had more than 3 missing days during the week, then the weekly average was not calculated and treated as missing data and excluded from the analysis. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Week 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage Change
  Erythema; Week 1; n= 38, 41, 39, 36, 38, 30: number analyzed (Participants) | 38 | 41 | 39 | 36 | 38 | 30
  Erythema; Week 1; n= 38, 41, 39, 36, 38, 30 | -25.9 (26.76) | -35.4 (37.86) | -17.1 (28.74) | -19.9 (27.26) | -19.3 (34.12) | -8.9 (37.07)
  Erythema; Week 2; n= 39, 39, 39, 38, 33, 30: number analyzed (Participants) | 39 | 39 | 39 | 38 | 33 | 30
  Erythema; Week 2; n= 39, 39, 39, 38, 33, 30 | -49.6 (34.30) | -49.1 (35.86) | -35.5 (33.15) | -36.0 (36.46) | -26.3 (39.75) | -12.8 (56.34)
  Erythema; Week 4; n= 38, 39, 38, 38, 30, 30: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 30
  Erythema; Week 4; n= 38, 39, 38, 38, 30, 30 | -51.3 (32.74) | -59.0 (32.86) | -55.7 (34.28) | -45.6 (38.10) | -33.3 (37.14) | -30.6 (42.23)
  Erythema; Week 8; n= 36, 37, 34, 37, 29, 25: number analyzed (Participants) | 36 | 37 | 34 | 37 | 29 | 25
  Erythema; Week 8; n= 36, 37, 34, 37, 29, 25 | -58.8 (31.24) | -69.8 (33.06) | -65.7 (26.89) | -58.6 (35.05) | -55.2 (40.36) | -44.0 (48.80)
  Erythema; Week 12; n= 36, 37, 32, 34, 28, 23: number analyzed (Participants) | 36 | 37 | 32 | 34 | 28 | 23
  Erythema; Week 12; n= 36, 37, 32, 34, 28, 23 | -69.9 (36.69) | -69.4 (37.37) | -77.1 (25.66) | -66.7 (34.33) | -51.2 (36.55) | -52.2 (38.70)
  Erythema; Week 14; n= 34, 35, 31, 32, 27, 23: number analyzed (Participants) | 34 | 35 | 31 | 32 | 27 | 23
  Erythema; Week 14; n= 34, 35, 31, 32, 27, 23 | -70.6 (36.71) | -66.2 (37.37) | -55.9 (46.66) | -49.5 (34.26) | -56.2 (35.55) | -48.6 (34.05)
  Erythema; Week 16; n= 34, 36 , 31, 34, 27, 23: number analyzed (Participants) | 34 | 36 | 31 | 34 | 27 | 23
  Erythema; Week 16; n= 34, 36 , 31, 34, 27, 23 | -67.2 (36.58) | -59.7 (39.11) | -60.2 (44.03) | -58.8 (36.29) | -50.6 (40.95) | -50.0 (30.57)
  Erythema; EW; n= 3, 4, 7, 3, 11, 11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  Erythema; EW; n= 3, 4, 7, 3, 11, 11 | -33.3 (57.74) | -8.3 (44.10) | -21.4 (48.80) | -50.0 (50.00) | -10.6 (42.99) | 18.2 (87.39)
  Induration/Papulation;Week 1; n=38,40,37,37,38,32: number analyzed (Participants) | 38 | 40 | 37 | 37 | 38 | 32
  Induration/Papulation;Week 1; n=38,40,37,37,38,32 | -18.0 (26.67) | -28.3 (33.16) | -21.6 (26.02) | -18.0 (25.27) | -12.7 (41.27) | -3.1 (35.78)
  Induration/Papulation;Week 2;n= 39,38,37,39,33,32: number analyzed (Participants) | 39 | 38 | 37 | 39 | 33 | 32
  Induration/Papulation;Week 2;n= 39,38,37,39,33,32 | -43.2 (40.05) | -46.9 (38.91) | -41.0 (40.37) | -40.6 (43.05) | -22.7 (47.47) | -14.6 (55.48)
  Induration/Papulation;Week 4;n= 38,38,36,39,30,32: number analyzed (Participants) | 38 | 38 | 36 | 39 | 30 | 32
  Induration/Papulation;Week 4;n= 38,38,36,39,30,32 | -49.1 (45.84) | -61.0 (38.22) | -56.5 (32.68) | -43.6 (51.24) | -31.1 (32.38) | -31.8 (43.04)
  Induration/Papulation;Week 8;n= 36,36,33,38,29,27: number analyzed (Participants) | 36 | 36 | 33 | 38 | 29 | 27
  Induration/Papulation;Week 8;n= 36,36,33,38,29,27 | -57.9 (35.07) | -58.8 (43.37) | -70.7 (27.96) | -65.8 (36.55) | -54.0 (46.64) | -44.4 (43.85)
  Induration/Papulation;Week 12;n=36,36,31,35,28,25: number analyzed (Participants) | 36 | 36 | 31 | 35 | 28 | 25
  Induration/Papulation;Week 12;n=36,36,31,35,28,25 | -72.2 (46.97) | -68.5 (43.60) | -79.6 (26.77) | -65.2 (34.39) | -41.7 (47.90) | -54.7 (40.69)
  Induration/Papulation;Week 14;n=34,34,30,33,27,25: number analyzed (Participants) | 34 | 34 | 30 | 33 | 27 | 25
  Induration/Papulation;Week 14;n=34,34,30,33,27,25 | -65.7 (44.18) | -73.5 (31.55) | -63.9 (32.48) | -46.5 (39.69) | -50.0 (48.48) | -56.0 (39.35)
  Induration/Papulation;Week 16;n=34,35,30,35,27,25: number analyzed (Participants) | 34 | 35 | 30 | 35 | 27 | 25
  Induration/Papulation;Week 16;n=34,35,30,35,27,25 | -65.7 (42.43) | -62.4 (38.84) | -67.8 (35.81) | -61.0 (38.97) | -51.2 (43.10) | -52.0 (49.14)
  Induration/Papulation; EW; n= 3,4,6,3,11,11: number analyzed (Participants) | 3 | 4 | 6 | 3 | 11 | 11
  Induration/Papulation; EW; n= 3,4,6,3,11,11 | 0.0 (100.00) | -12.5 (62.92) | -16.7 (68.31) | 0.0 (100.00) | -4.5 (56.81) | 27.3 (103.35)
  Lichenification; Week 1;n=34,37,38,37,37,32: number analyzed (Participants) | 34 | 37 | 38 | 37 | 37 | 32
  Lichenification; Week 1;n=34,37,38,37,37,32 | -22.1 (39.51) | -30.6 (40.73) | -24.6 (39.85) | -16.7 (33.10) | -19.8 (29.88) | -13.5 (28.54)
  Lichenification; Week 2;n=35,36,38,39,32,32: number analyzed (Participants) | 35 | 36 | 38 | 39 | 32 | 32
  Lichenification; Week 2;n=35,36,38,39,32,32 | -38.1 (45.83) | -46.3 (42.56) | -36.8 (37.60) | -38.5 (41.56) | -39.1 (39.85) | -19.3 (46.97)
  Lichenification; Week 4;n=34,36,37,39,29,32: number analyzed (Participants) | 34 | 36 | 37 | 39 | 29 | 32
  Lichenification; Week 4;n=34,36,37,39,29,32 | -47.1 (48.80) | -51.9 (36.47) | -56.3 (37.34) | -45.3 (40.64) | -32.2 (46.91) | -23.4 (48.61)
  Lichenification; Week 8;n=33,35,33,38,28,27: number analyzed (Participants) | 33 | 35 | 33 | 38 | 28 | 27
  Lichenification; Week 8;n=33,35,33,38,28,27 | -53.5 (47.10) | -62.9 (38.58) | -62.1 (32.62) | -60.1 (39.24) | -53.0 (36.59) | -49.4 (37.12)
  Lichenification; Week 12;n=33,35,31,35,27,25: number analyzed (Participants) | 33 | 35 | 31 | 35 | 27 | 25
  Lichenification; Week 12;n=33,35,31,35,27,25 | -71.7 (41.56) | -69.0 (36.86) | -78.5 (23.25) | -64.8 (37.44) | -57.4 (36.50) | -67.3 (35.84)
  Lichenification; Week 14;n=31,33,30,33,26,25: number analyzed (Participants) | 31 | 33 | 30 | 33 | 26 | 25
  Lichenification; Week 14;n=31,33,30,33,26,25 | -73.7 (38.19) | -62.6 (43.71) | -59.4 (43.92) | -56.6 (36.07) | -54.5 (40.15) | -60.7 (36.92)
  Lichenification; Week 16;n=31,34,30,35,26,25: number analyzed (Participants) | 31 | 34 | 30 | 35 | 26 | 25
  Lichenification; Week 16;n=31,34,30,35,26,25 | -65.6 (45.12) | -60.3 (43.81) | -66.1 (34.04) | -60.0 (37.31) | -57.7 (39.79) | -68.7 (33.44)
  Lichenification; EW;n= 2,2,7,3,11,11: number analyzed (Participants) | 2 | 2 | 7 | 3 | 11 | 11
  Lichenification; EW;n= 2,2,7,3,11,11 | -50.0 (70.71) | -25.0 (106.07) | -21.4 (69.86) | -50.0 (50.00) | -16.7 (39.44) | -9.1 (62.52)
  Oozing/crusting; Week 1;n=24,21,26,27,27,22: number analyzed (Participants) | 24 | 21 | 26 | 27 | 27 | 22
  Oozing/crusting; Week 1;n=24,21,26,27,27,22 | -29.2 (52.99) | -61.9 (47.18) | -40.4 (46.95) | -40.7 (48.11) | -44.4 (65.54) | -20.5 (50.38)
  Oozing/crusting; Week 2;n=24,21,27,28,22,23: number analyzed (Participants) | 24 | 21 | 27 | 28 | 22 | 23
  Oozing/crusting; Week 2;n=24,21,27,28,22,23 | -64.6 (47.73) | -64.3 (42.26) | -75.9 (37.65) | -51.8 (48.08) | -62.9 (44.52) | -37.0 (43.22)
  Oozing/crusting; Week 4;n= 24,21,27,28,21,24: number analyzed (Participants) | 24 | 21 | 27 | 28 | 21 | 24
  Oozing/crusting; Week 4;n= 24,21,27,28,21,24 | -75.0 (44.23) | -69.0 (43.23) | -79.0 (44.96) | -76.8 (41.90) | -68.3 (43.75) | -45.8 (55.00)
  Oozing/crusting; Week 8;n=23,20,25,27,21,21: number analyzed (Participants) | 23 | 20 | 25 | 27 | 21 | 21
  Oozing/crusting; Week 8;n=23,20,25,27,21,21 | -82.6 (38.76) | -97.5 (11.18) | -84.7 (33.99) | -85.2 (36.20) | -65.9 (43.29) | -59.5 (56.17)
  Oozing/crusting; Week 12;n=23,20,23,25,21,19: number analyzed (Participants) | 23 | 20 | 23 | 25 | 21 | 19
  Oozing/crusting; Week 12;n=23,20,23,25,21,19 | -84.8 (35.15) | -87.5 (31.93) | -97.8 (10.43) | -86.0 (33.91) | -74.6 (40.35) | -73.7 (71.43)
  Oozing/crusting; Week 14;n=22,19,23,23,21,19: number analyzed (Participants) | 22 | 19 | 23 | 23 | 21 | 19
  Oozing/crusting; Week 14;n=22,19,23,23,21,19 | -86.4 (35.13) | -73.7 (56.20) | -84.8 (32.14) | -80.4 (39.14) | -84.9 (33.29) | -76.3 (42.06)
  Oozing/crusting; Week 16;n=22,20,23,25,21,19: number analyzed (Participants) | 22 | 20 | 23 | 25 | 21 | 19
  Oozing/crusting; Week 16;n=22,20,23,25,21,19 | -79.5 (39.82) | -80.0 (41.04) | -84.8 (35.15) | -84.0 (34.52) | -75.4 (41.37) | -71.1 (56.06)
  Oozing/crusting; EW;n=1,1,4,2,5,5: number analyzed (Participants) | 1 | 1 | 4 | 2 | 5 | 5
  Oozing/crusting; EW;n=1,1,4,2,5,5 | -100.0 (NA) — NA indicates that data is not available | 0.0 (NA) — NA indicates that data is not available | -12.5 (103.08) | 0.0 (0.00) | -20.0 (44.72) | -20.0 (44.72)
  Scaling; Week 1;n=34,36,34,35,36,29: number analyzed (Participants) | 34 | 36 | 34 | 35 | 36 | 29
  Scaling; Week 1;n=34,36,34,35,36,29 | -28.4 (52.79) | -36.1 (47.22) | -32.8 (47.76) | -19.5 (58.23) | -24.1 (41.87) | -8.6 (42.40)
  Scaling; Week 2;n= 35,34,34,37,31,30: number analyzed (Participants) | 35 | 34 | 34 | 37 | 31 | 30
  Scaling; Week 2;n= 35,34,34,37,31,30 | -47.1 (45.28) | -64.7 (45.28) | -53.4 (42.60) | -44.1 (51.10) | -36.6 (40.69) | -12.8 (43.04)
  Scaling; Week 4;n=35,34,34,37,28,30: number analyzed (Participants) | 35 | 34 | 34 | 37 | 28 | 30
  Scaling; Week 4;n=35,34,34,37,28,30 | -57.1 (45.61) | -69.1 (40.85) | -68.1 (47.38) | -51.8 (52.08) | -38.1 (36.81) | -33.3 (53.07)
  Scaling; Week 8;n=33,32,30,36,27,25: number analyzed (Participants) | 33 | 32 | 30 | 36 | 27 | 25
  Scaling; Week 8;n=33,32,30,36,27,25 | -57.6 (50.19) | -81.3 (35.36) | -81.7 (30.75) | -67.1 (43.00) | -59.3 (38.49) | -50.0 (52.04)
  Scaling; Week 12;n=33,32,29,33,26,23: number analyzed (Participants) | 33 | 32 | 29 | 33 | 26 | 23
  Scaling; Week 12;n=33,32,29,33,26,23 | -75.8 (41.69) | -84.4 (32.22) | -82.8 (30.69) | -71.2 (48.46) | -64.7 (37.51) | -54.3 (52.03)
  Scaling; Week 14;n=31,30,28,31,25,23: number analyzed (Participants) | 31 | 30 | 28 | 31 | 25 | 23
  Scaling; Week 14;n=31,30,28,31,25,23 | -74.2 (40.56) | -73.3 (48.66) | -70.2 (39.11) | -60.2 (63.78) | -62.0 (39.24) | -52.2 (43.90)
  Scaling; Week 16;n=31,31,28,33,25,23: number analyzed (Participants) | 31 | 31 | 28 | 33 | 25 | 23
  Scaling; Week 16;n=31,31,28,33,25,23 | -75.8 (48.08) | -66.1 (50.64) | -72.0 (36.87) | -65.7 (44.08) | -70.7 (35.45) | -51.4 (51.23)
  Scaling; EW;n=2,4,5,3,9,9: number analyzed (Participants) | 2 | 4 | 5 | 3 | 9 | 9
  Scaling; EW;n=2,4,5,3,9,9 | -50.0 (70.71) | 0.0 (141.42) | -10.0 (74.16) | -50.0 (50.00) | -5.6 (76.83) | 0.0 (70.71)

15. Secondary Outcome: Mean Change From Baseline in Body Surface Area (Percent BSA)
Description: The extent of BSA affected by AD is a general indicator of disease severity and the assessment of BSA with AD was performed separately for four body surface regions: the head (h), the upper extremities (u), the trunk (t) and the lower extremities (l), corresponding to 10, 20, 30, and 40 percent of the total body area, respectively. Mean change from Baseline in percent BSA was presented using mean and SD at Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and EW visit. Baseline was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage of surface area
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage of surface area
  Week 1; n= 38, 41, 39, 37, 38, 32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38, 41, 39, 37, 38, 32 | -2.37 (4.774) | -3.57 (5.498) | -2.44 (4.313) | -1.52 (6.078) | -0.33 (6.591) | -0.25 (4.411)
  Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39, 39, 39, 39, 33, 32 | -4.99 (7.330) | -7.07 (6.639) | -4.88 (5.243) | -3.78 (5.897) | -2.01 (6.484) | -0.04 (4.698)
  Week 4; n= 38, 39, 38, 39, 30, 32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38, 39, 38, 39, 30, 32 | -7.37 (6.276) | -9.76 (8.581) | -7.47 (7.567) | -7.07 (6.382) | -2.93 (7.772) | -2.05 (6.517)
  Week 8; n= 36, 37, 34, 38, 29, 27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36, 37, 34, 38, 29, 27 | -9.23 (8.425) | -11.70 (9.208) | -10.89 (9.692) | -8.56 (6.217) | -5.41 (7.961) | -3.33 (7.264)
  Week 12; n= 36, 37, 32, 35, 28, 25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36, 37, 32, 35, 28, 25 | -11.19 (8.643) | -11.55 (9.690) | -12.18 (9.581) | -9.81 (7.717) | -6.00 (8.424) | -5.44 (8.079)
  Week 14; n= 34, 35, 31, 33, 27, 25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34, 35, 31, 33, 27, 25 | -9.25 (7.121) | -9.85 (9.446) | -11.26 (10.262) | -9.26 (7.529) | -5.60 (7.575) | -5.80 (6.987)
  Week 16; n= 34, 36, 31, 35, 27, 25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34, 36, 31, 35, 27, 25 | -8.19 (7.826) | -9.93 (8.820) | -10.92 (9.903) | -9.25 (8.399) | -5.66 (7.695) | -5.53 (7.227)
  EW; n= 3, 4, 7, 3, 11, 11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3, 4, 7, 3, 11, 11 | -2.60 (4.613) | 4.63 (9.586) | 5.36 (21.468) | 3.20 (14.468) | 3.36 (9.492) | 7.50 (18.476)

16. Secondary Outcome: Mean Change From Baseline in IGA Score
Description: The IGA is a clinical tool for assessing the current state/severity of a participant's AD. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines. IGA is made without reference to previous scores. Score ranges from 0 (clear) to 4 (severe). Higher values represent a severe disease. Mean change from Baseline in IGA score was presented using mean and SD at Week 1, Week 2, Week 4, Week 8, Week 12, Week 14 (follow up 1), Week 16 (follow up 2) and EW visit. Baseline was defined as the latest assessment prior to first dose and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to Week 16)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Scores on a scale
  Week 1; n= 38, 41, 39, 37, 38, 32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38, 41, 39, 37, 38, 32 | -0.5 (0.60) | -0.6 (0.67) | -0.3 (0.48) | -0.4 (0.55) | -0.3 (0.58) | -0.4 (0.62)
  Week 2; n= 39, 39, 39, 39, 33, 32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39, 39, 39, 39, 33, 32 | -1.0 (0.69) | -0.9 (0.70) | -0.6 (0.67) | -0.7 (0.79) | -0.7 (0.72) | -0.5 (0.72)
  Week 4; n= 38, 39, 38, 39, 30, 32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38, 39, 38, 39, 30, 32 | -1.3 (0.86) | -1.4 (0.81) | -1.1 (0.77) | -1.0 (0.81) | -1.0 (0.72) | -0.7 (0.82)
  Week 8; n= 36, 37, 34, 38, 29, 27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36, 37, 34, 38, 29, 27 | -1.4 (0.83) | -1.6 (0.82) | -1.3 (0.84) | -1.4 (0.85) | -1.2 (0.60) | -1.0 (0.88)
  Week 12; n= 36, 37, 32, 35, 28, 25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36, 37, 32, 35, 28, 25 | -1.7 (0.96) | -1.6 (0.83) | -1.6 (0.76) | -1.5 (0.95) | -1.3 (0.72) | -1.2 (0.78)
  Week 14; n= 34, 35, 31, 33, 27, 25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34, 35, 31, 33, 27, 25 | -1.5 (1.08) | -1.4 (0.77) | -1.5 (0.99) | -1.3 (0.92) | -1.2 (0.85) | -1.2 (0.75)
  Week 16; n= 34, 36, 31, 35, 27, 25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34, 36, 31, 35, 27, 25 | -1.2 (1.07) | -1.2 (0.74) | -1.4 (0.91) | -1.3 (0.94) | -1.3 (0.90) | -1.1 (0.73)
  EW; n= 3, 4, 7, 3, 11, 11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3, 4, 7, 3, 11, 11 | -1.3 (1.53) | 0.3 (0.50) | -0.6 (0.98) | -1.0 (1.00) | 0.1 (0.30) | 0.0 (0.89)

17. Secondary Outcome: Percentage of Participants Who Have an IGA Score of Clear or Almost Clear (0 or 1) and a Minimum 2 Grade Improvement in IGA Score From Baseline to Each Study Visit
Description: The IGA is a clinical tool for assessing the current state/severity of a participant's AD. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines. IGA is made without reference to previous scores. The percentage of participants who have an IGA score of clear or almost clear and a minimum 2 grade improvement from Baseline to each study visit in IGA score was presented. The statistical analysis was performed using a repeated measures factorial logistic regression model with covariates for dose, frequency of administration, and study day as well as a dose by frequency interaction term. The analysis was performed on ITT Population which comprised of all randomized participants. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category title).
Time Frame: Weeks 1, 2, 4, 8, 12, 14, 16, EW (up to week 16)
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Percentage of participants
  Week 1; n= 38,41,39,37,38,32: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 32
  Week 1; n= 38,41,39,37,38,32 | 5 | 5 | 0 | 3 | 3 | 3
  Week 2; n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39,39,39,39,33,32 | 18 | 18 | 10 | 13 | 15 | 9
  Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38,39,38,39,30,32 | 32 | 38 | 26 | 23 | 20 | 9
  Week 8; n= 36,37,34,38,29,27: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 27
  Week 8; n= 36,37,34,38,29,27 | 42 | 54 | 38 | 42 | 28 | 19
  Week 12; n= 36,37,32,35,28,25: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 25
  Week 12; n= 36,37,32,35,28,25 | 58 | 51 | 50 | 40 | 36 | 44
  Week 14; n= 34,35,31,33,27,25: number analyzed (Participants) | 34 | 35 | 31 | 33 | 27 | 25
  Week 14; n= 34,35,31,33,27,25 | 44 | 43 | 52 | 36 | 26 | 36
  Week 16; n= 34,36,31,35,27,25: number analyzed (Participants) | 34 | 36 | 31 | 35 | 27 | 25
  Week 16; n= 34,36,31,35,27,25 | 35 | 36 | 39 | 40 | 30 | 28
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | 33 | 0 | 14 | 33 | 0 | 9
Statistical Analysis 1: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = -7.7, 95% CI 2-sided [-45.8 to 32.5] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 1 has been presented
Statistical Analysis 2: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 15.4, 95% CI 2-sided [-25.7 to 52.6] — Difference between GSK2894512 1 % QD and vehicle QD at Week 1 has been presented
Statistical Analysis 3: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = -7.7, 95% CI 2-sided [-46.0 to 32.6] — Difference between GSK2894512 0.5 % BID and vehicle BID at Week 1 has been presented
Statistical Analysis 4: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 9.1, 95% CI 2-sided [-32.2 to 48.8] — Difference between GSK2894512 0.5 % QD and vehicle QD at Week 1 has been presented
Statistical Analysis 5: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = -24.2, 95% CI 2-sided [-60.8 to 14.8] — Difference between GSK2894512 1 % BID and vehicle BID at Week 2 has been presented
Statistical Analysis 6: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 28.5, 95% CI 2-sided [-13.7 to 63.0] — Difference between GSK2894512 1 % QD and vehicle QD at Week 2 has been presented
Statistical Analysis 7: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = -33.3, 95% CI 2-sided [-67.4 to 6.1] — Difference between GSK2894512 0.5 % BID and vehicle BID at Week 2 has been presented
Statistical Analysis 8: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = -0.9, 95% CI 2-sided [-40.7 to 40.7] — Difference between GSK2894512 0.5 % QD and vehicle QD at Week 2 has been presented
Statistical Analysis 9: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = -15.2, 95% CI 2-sided [-53.8 to 23.5] — Difference between GSK2894512 1 % BID and vehicle BID at Week 4 has been presented
Statistical Analysis 10: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 43.4, 95% CI 2-sided [2.7 to 74.6] — Difference between GSK2894512 1 % QD and vehicle QD at Week 4 has been presented
Statistical Analysis 11: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = -15.2, 95% CI 2-sided [-53.8 to 23.5] — Difference between GSK2894512 0.5 % BID and vehicle BID at Week 4 has been presented
Statistical Analysis 12: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 9.1, 95% CI 2-sided [-35.6 to 51.2] — Difference between GSK2894512 0.5 % QD and vehicle QD at Week 4 has been presented
Statistical Analysis 13: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 18.3, 95% CI 2-sided [-25.1 to 57.1] — Difference between GSK2894512 1 % BID and vehicle BID at Week 8 has been presented
Statistical Analysis 14: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 47.7, 95% CI 2-sided [4.8 to 78.7] — Difference between GSK2894512 1 % QD and vehicle QD at Week 8 has been presented
Statistical Analysis 15: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = -11.7, 95% CI 2-sided [-51.3 to 30.2] — Difference between GSK2894512 0.5 % BID and vehicle BID at Week 8 has been presented
Statistical Analysis 16: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = 9.1, 95% CI 2-sided [-35.6 to 51.2] — Difference between GSK2894512 0.5 % QD and vehicle QD at Week 8 has been presented
Statistical Analysis 17: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = 6.4, 95% CI 2-sided [-35.4 to 48.5] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 18: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 6.0, 95% CI 2-sided [-35.8 to 47.1] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 19: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = -13.6, 95% CI 2-sided [-54.0 to 31.2] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 20: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = -25.6, 95% CI 2-sided [-65.3 to 22.4] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 21: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = -1.0, 95% CI 2-sided [-44.5 to 42.7] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 22: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 5.6, 95% CI 2-sided [-37.8 to 47.3] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 23: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = -5.5, 95% CI 2-sided [-47.9 to 37.6] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 24: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Difference in percentages = -4.4, 95% CI 2-sided [-48.3 to 41.5] — Difference between GSK2894512 0.5 % QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 25: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Difference in percentages = -1.0, 95% CI 2-sided [-44.5 to 42.7] — Difference between GSK2894512 1 % BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 26: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Difference in percentages = 8.3, 95% CI 2-sided [-35.0 to 49.2] — Difference between GSK2894512 1 % QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 27: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Difference in percentages = -3.3, 95% CI 2-sided [-46.0 to 42.3] — Difference between GSK2894512 0.5 % BID and Vehicle BID at Week 16 has been presented

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function. Treatment emergent AEs (TEAE) is defined as AE occurred on or after study treatment start date and on or before last visit. Number of participants with AEs and serious TEAEs were presented. The analysis was performed on Safety population which comprised of all participants who receive at least one dose of study treatment.
Time Frame: Weeks 1, 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  TEAEs | 28 | 22 | 20 | 23 | 19 | 15
  Serious TEAEs | 1 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Reported Tolerability Score of 0 to 4 Over Time
Description: Participants were asked to use a 5-point tolerability scale from 0 (none) to 4 (severe) to assess the presence and degree of burning/stinging and itching at the application sites that has generally been experienced following application of the study treatment. The score represented an 'average' across all application sites. A score of 3 or 4 was reported as an AE. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Week 1, 2, 4, 8, 12, 14, EW (up to Week 14)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  Week 1; none; n= 38,40,39,37,38,33: number analyzed (Participants) | 38 | 40 | 39 | 37 | 38 | 33
  Week 1; none; n= 38,40,39,37,38,33 | 19 | 25 | 25 | 21 | 15 | 22
  Week 1; slight; n= 38,40,39,37,38,33: number analyzed (Participants) | 38 | 40 | 39 | 37 | 38 | 33
  Week 1; slight; n= 38,40,39,37,38,33 | 6 | 10 | 5 | 6 | 9 | 5
  Week 1; mild; n= 38,40,39,37,38,33: number analyzed (Participants) | 38 | 40 | 39 | 37 | 38 | 33
  Week 1; mild; n= 38,40,39,37,38,33 | 9 | 3 | 2 | 8 | 6 | 3
  Week 1; Moderate; n= 38,40,39,37,38,33: number analyzed (Participants) | 38 | 40 | 39 | 37 | 38 | 33
  Week 1; Moderate; n= 38,40,39,37,38,33 | 2 | 2 | 6 | 2 | 7 | 2
  Week 1; severe; n= 38,40,39,37,38,33: number analyzed (Participants) | 38 | 40 | 39 | 37 | 38 | 33
  Week 1; severe; n= 38,40,39,37,38,33 | 2 | 0 | 1 | 0 | 1 | 1
  Week 2; none; n= 39,37,39,39,33,32: number analyzed (Participants) | 39 | 37 | 39 | 39 | 33 | 32
  Week 2; none; n= 39,37,39,39,33,32 | 26 | 27 | 33 | 20 | 16 | 18
  Week 2; slight;n= 39,37,39,39,33,32: number analyzed (Participants) | 39 | 37 | 39 | 39 | 33 | 32
  Week 2; slight;n= 39,37,39,39,33,32 | 5 | 5 | 1 | 11 | 6 | 5
  Week 2; mild; n= 39,37,39,39,33,32: number analyzed (Participants) | 39 | 37 | 39 | 39 | 33 | 32
  Week 2; mild; n= 39,37,39,39,33,32 | 3 | 4 | 4 | 4 | 8 | 5
  Week 2; moderate; n= 39,37,39,39,33,32: number analyzed (Participants) | 39 | 37 | 39 | 39 | 33 | 32
  Week 2; moderate; n= 39,37,39,39,33,32 | 4 | 0 | 1 | 3 | 2 | 2
  Week 2; severe; n= 39,37,39,39,33,32: number analyzed (Participants) | 39 | 37 | 39 | 39 | 33 | 32
  Week 2; severe; n= 39,37,39,39,33,32 | 1 | 1 | 0 | 1 | 1 | 2
  Week 4; none; n= 38, 39, 38,39,29,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 29 | 32
  Week 4; none; n= 38, 39, 38,39,29,32 | 26 | 26 | 27 | 27 | 15 | 21
  Week 4; slight; n= 38, 39, 38,39,29,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 29 | 32
  Week 4; slight; n= 38, 39, 38,39,29,32 | 7 | 8 | 5 | 9 | 8 | 2
  Week 4; mild; n= 38, 39, 38,39,29,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 29 | 32
  Week 4; mild; n= 38, 39, 38,39,29,32 | 3 | 4 | 6 | 2 | 4 | 5
  Week 4; moderate; n= 38, 39, 38,39,29,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 29 | 32
  Week 4; moderate; n= 38, 39, 38,39,29,32 | 2 | 1 | 0 | 1 | 2 | 3
  Week 4; severe; n= 38, 39, 38,39,29,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 29 | 32
  Week 4; severe; n= 38, 39, 38,39,29,32 | 0 | 0 | 0 | 0 | 0 | 1
  Week 8; none; n= 36, 37, 34, 38, 29, 28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Week 8; none; n= 36, 37, 34, 38, 29, 28 | 25 | 28 | 23 | 29 | 19 | 17
  Week 8; slight; n= 36, 37, 34, 38, 29, 28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Week 8; slight; n= 36, 37, 34, 38, 29, 28 | 6 | 6 | 8 | 7 | 5 | 5
  Week 8; mild; n= 36, 37, 34, 38, 29, 28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Week 8; mild; n= 36, 37, 34, 38, 29, 28 | 3 | 2 | 2 | 2 | 3 | 3
  Week 8; moderate; n= 36, 37, 34, 38, 29, 28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Week 8; moderate; n= 36, 37, 34, 38, 29, 28 | 1 | 1 | 1 | 0 | 1 | 3
  Week 8; severe; n= 36, 37, 34, 38, 29, 28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Week 8; severe; n= 36, 37, 34, 38, 29, 28 | 1 | 0 | 0 | 0 | 1 | 0
  Week 12; none; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; none; n= 36, 37, 32, 35, 28, 28 | 24 | 27 | 26 | 27 | 16 | 23
  Week 12; slight; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; slight; n= 36, 37, 32, 35, 28, 28 | 6 | 8 | 3 | 6 | 8 | 3
  Week 12; mild; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; mild; n= 36, 37, 32, 35, 28, 28 | 5 | 1 | 3 | 2 | 3 | 0
  Week 12; moderate; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; moderate; n= 36, 37, 32, 35, 28, 28 | 1 | 0 | 0 | 0 | 1 | 0
  Week 12; severe; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; severe; n= 36, 37, 32, 35, 28, 28 | 0 | 1 | 0 | 0 | 0 | 2
  Week 14; none; n= 34,35,32,33,31,29: number analyzed (Participants) | 34 | 35 | 32 | 33 | 31 | 29
  Week 14; none; n= 34,35,32,33,31,29 | 26 | 29 | 27 | 26 | 22 | 22
  Week 14; slight; n= 34,35,32,33,31,29: number analyzed (Participants) | 34 | 35 | 32 | 33 | 31 | 29
  Week 14; slight; n= 34,35,32,33,31,29 | 4 | 5 | 4 | 5 | 4 | 4
  Week 14; mild; n= 34,35,32,33,31,29: number analyzed (Participants) | 34 | 35 | 32 | 33 | 31 | 29
  Week 14; mild; n= 34,35,32,33,31,29 | 3 | 0 | 0 | 2 | 2 | 2
  Week 14; moderate; n= 34,35,32,33,31,29: number analyzed (Participants) | 34 | 35 | 32 | 33 | 31 | 29
  Week 14; moderate; n= 34,35,32,33,31,29 | 1 | 1 | 1 | 0 | 2 | 1
  Week 14; severe; n= 34,35,32,33,31,29: number analyzed (Participants) | 34 | 35 | 32 | 33 | 31 | 29
  Week 14; severe; n= 34,35,32,33,31,29 | 0 | 0 | 0 | 0 | 1 | 0
  EW; none; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; none; n= 3,4,7,3,11,11 | 2 | 1 | 4 | 2 | 3 | 7
  EW; slight; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; slight; n= 3,4,7,3,11,11 | 0 | 1 | 0 | 0 | 4 | 0
  EW; mild; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; mild; n= 3,4,7,3,11,11 | 1 | 1 | 0 | 0 | 0 | 1
  EW; moderate; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; moderate; n= 3,4,7,3,11,11 | 0 | 1 | 2 | 1 | 1 | 2
  EW; severe; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; severe; n= 3,4,7,3,11,11 | 0 | 0 | 1 | 0 | 3 | 1

20. Secondary Outcome: Change From Baseline in Albumin and Total Protein
Description: Blood samples were collected to evaluate change from Baseline in albumin and total protein values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 1, 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Gram per Liter (G/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Gram per Liter (G/L)
  Albumin; Week 2; n=38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Albumin; Week 2; n=38,39,38,39,33,32 | -1.2 (2.96) | -1.3 (1.89) | -2.2 (2.96) | -1.4 (2.02) | -1.2 (3.91) | -1.2 (2.17)
  Albumin; Week 4; n=38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Albumin; Week 4; n=38,39,38,38,30,32 | -1.1 (2.87) | -0.6 (2.17) | -1.9 (2.49) | -1.3 (2.74) | -1.2 (2.46) | -0.7 (2.74)
  Albumin; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Albumin; Week 8; n= 35,37,34,38,29,28 | -1.7 (2.47) | -1.0 (1.86) | -1.9 (2.38) | -1.1 (2.29) | -1.4 (2.54) | -1.4 (3.14)
  Albumin; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Albumin; Week 12; n= 36,37,32,35,28,28 | -1.1 (2.48) | -1.2 (2.65) | -2.2 (2.35) | -1.7 (2.47) | -1.6 (2.79) | -0.9 (2.09)
  Albumin; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Albumin; Week 14; n= 33,35,32,34,31,29 | -1.6 (2.36) | -1.5 (2.41) | -2.0 (2.48) | -1.6 (3.04) | -2.0 (2.70) | -0.9 (2.21)
  Albumin; EW;n = 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Albumin; EW;n = 3,3,7,3,11,11 | -1.3 (4.04) | -3.3 (2.52) | -3.0 (1.29) | -0.7 (0.58) | -0.7 (2.87) | -2.5 (2.84)
  Total protein; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Total protein; Week 2; n= 38,39,38,39,33,32 | -1.5 (4.49) | -2.2 (2.84) | -2.3 (4.48) | -2.0 (3.34) | -1.9 (6.66) | -1.6 (3.31)
  Total protein; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Total protein; Week 4; n= 38,39,38,38,30,32 | -1.9 (4.32) | -1.1 (3.49) | -2.4 (4.43) | -1.7 (5.12) | -2.3 (3.86) | -1.1 (4.62)
  Total protein; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Total protein; Week 8; n= 35,37,34,38,29,28 | -2.8 (3.91) | -2.1 (3.02) | -2.8 (4.46) | -1.7 (3.89) | -1.7 (4.09) | -1.8 (4.82)
  Total protein; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Total protein; Week 12; n= 36,37,32,35,28,28 | -2.0 (4.16) | -2.5 (4.43) | -3.8 (4.40) | -2.4 (4.07) | -2.2 (5.38) | -1.0 (3.18)
  Total protein; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Total protein; Week 14; n= 33,35,32,34,31,29 | -3.0 (3.80) | -2.4 (3.23) | -3.3 (4.07) | -2.0 (4.75) | -2.3 (4.26) | -1.3 (3.84)
  Total protein; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Total protein; EW; n= 3,3,7,3,11,11 | -2.3 (6.43) | -4.0 (2.00) | -2.0 (2.16) | -1.0 (2.00) | -1.4 (3.64) | -3.0 (5.08)

21. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (Alk.Phosph.), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Gamma Glutamyl Transferase (GGT)
Description: Blood samples were collected to evaluate change from Baseline in Alk.phosph., ALT, AST and GGT values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
International unit per liter (IU/L)
  Alk.Phosph.; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Alk.Phosph.; Week 2; n= 38,39,38,39,33,32 | 3.7 (14.58) | -1.7 (12.24) | 3.7 (21.04) | -2.3 (13.49) | -2.3 (15.32) | -2.0 (8.70)
  Alk.Phosph.; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Alk.Phosph.; Week 4; n= 38,39,38,38,30,32 | 2.1 (15.59) | -0.4 (12.17) | 1.7 (15.22) | -2.7 (12.36) | -3.8 (16.24) | -3.9 (9.79)
  Alk.Phosph.; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Alk.Phosph.; Week 8; n= 35,37,34,38,29,28 | 2.0 (12.40) | -0.7 (9.39) | -1.2 (12.85) | -4.8 (18.15) | -1.6 (19.08) | -5.7 (12.03)
  Alk.Phosph.; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Alk.Phosph.; Week 12; n= 36,37,32,35,28,28 | 3.1 (15.36) | -0.4 (10.14) | -5.1 (18.47) | -6.3 (17.29) | -8.1 (21.60) | -7.8 (15.34)
  Alk. Phosph.; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Alk. Phosph.; Week 14; n= 33,35,32,34,31,29 | -1.4 (13.46) | -3.0 (17.56) | -7.2 (19.31) | -7.2 (20.07) | -6.5 (24.86) | -8.3 (14.83)
  Alk.Phosph.; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Alk.Phosph.; EW; n= 3,3,7,3,11,11 | -2.3 (27.74) | 5.3 (12.50) | 8.0 (18.13) | 0.3 (9.87) | 0.9 (6.74) | -0.5 (7.39)
  ALT; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  ALT; Week 2; n= 38,39,38,39,33,32 | 3.6 (21.02) | -1.8 (3.92) | 7.7 (28.01) | 1.5 (12.52) | 0.2 (7.21) | 0.2 (6.06)
  ALT; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  ALT; Week 4; n= 38,39,38,38,30,32 | -0.8 (9.20) | -1.1 (5.23) | 2.7 (8.07) | 1.7 (9.28) | 0.3 (7.63) | 0.6 (4.55)
  ALT; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  ALT; Week 8; n= 35,37,34,38,29,28 | 4.9 (30.93) | -1.4 (7.00) | 1.2 (6.77) | -1.5 (3.98) | -2.0 (6.06) | 0.3 (5.16)
  ALT; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  ALT; Week 12; n= 36,37,32,35,28,28 | -0.3 (12.51) | -3.1 (4.78) | -1.4 (4.13) | -0.6 (4.64) | 0.8 (7.97) | -0.2 (5.58)
  ALT; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  ALT; Week 14; n= 33,35,32,34,31,29 | 3.3 (24.10) | -3.2 (5.47) | -0.9 (4.51) | -1.0 (3.93) | -0.5 (5.58) | -0.8 (3.15)
  ALT; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  ALT; EW; n= 3,3,7,3,11,11 | 13.0 (37.64) | -3.7 (16.62) | 11.3 (36.60) | 2.0 (6.56) | -1.7 (4.73) | 3.3 (7.70)
  AST; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  AST; Week 2; n= 38,39,38,39,33,32 | 1.6 (9.36) | -1.3 (2.98) | 3.1 (13.84) | 0.2 (4.99) | -0.8 (4.99) | 0.5 (3.54)
  AST; Week 4; n=38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  AST; Week 4; n=38,39,38,38,30,32 | -0.4 (5.24) | -1.1 (4.18) | 1.0 (6.37) | 1.1 (6.81) | 0.0 (5.68) | 0.5 (4.17)
  AST; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  AST; Week 8; n= 35,37,34,38,29,28 | 18.4 (97.92) | -0.9 (5.06) | 0.2 (4.80) | -1.1 (4.56) | -1.9 (6.05) | -0.1 (5.80)
  AST; Week 12; n=36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  AST; Week 12; n=36,37,32,35,28,28 | 0.1 (8.54) | -1.2 (4.67) | -1.3 (5.12) | -0.7 (4.90) | 0.9 (6.88) | 0.2 (5.20)
  AST; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  AST; Week 14; n= 33,35,32,34,31,29 | 4.4 (28.19) | -2.2 (4.89) | -1.3 (3.92) | -1.1 (3.48) | 0.5 (8.12) | 0.0 (4.49)
  AST; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  AST; EW; n= 3,3,7,3,11,11 | 4.7 (8.62) | 1.7 (14.57) | 4.0 (12.83) | 3.0 (1.73) | -0.8 (2.14) | 3.1 (6.30)
  GGT; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  GGT; Week 2; n= 38,39,38,39,33,32 | -0.3 (6.36) | -1.3 (4.61) | 4.0 (13.82) | 0.7 (3.49) | -0.9 (8.04) | -2.9 (9.86)
  GGT; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  GGT; Week 4; n= 38,39,38,38,30,32 | -2.1 (9.47) | -0.8 (4.01) | 1.3 (6.38) | 0.9 (4.87) | 0.1 (10.95) | -1.0 (4.79)
  GGT; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  GGT; Week 8; n= 35,37,34,38,29,28 | -2.0 (14.19) | -1.2 (4.80) | 1.6 (10.32) | -0.5 (6.96) | -0.2 (11.68) | 0.4 (5.73)
  GGT; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  GGT; Week 12; n= 36,37,32,35,28,28 | -1.8 (14.77) | -1.6 (4.05) | 0.8 (8.38) | 1.1 (4.52) | 1.7 (11.65) | 1.9 (7.12)
  GGT; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  GGT; Week 14; n= 33,35,32,34,31,29 | -2.2 (15.76) | -1.0 (3.43) | 0.7 (4.93) | 1.0 (3.63) | 0.1 (8.19) | -0.3 (3.07)
  GGT; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  GGT; EW; n= 3,3,7,3,11,11 | 5.7 (31.01) | -8.0 (16.52) | 3.7 (9.48) | -0.7 (7.23) | -1.9 (8.19) | -4.8 (17.11)

22. Secondary Outcome: Change From Baseline in Direct and Total Bilirubin, Creatinine and Urate
Description: Blood samples were collected to evaluate change from Baseline in direct and total bilirubin, creatinine and urate values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Micromoles per liter (µmol/L)
  Direct bilirubin; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Direct bilirubin; Week 2; n= 38,39,38,39,33,32 | -0.1 (0.98) | -0.3 (1.08) | -0.5 (1.18) | -0.1 (1.07) | 0.0 (1.66) | -0.3 (1.15)
  Direct bilirubin; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Direct bilirubin; Week 4; n= 38,39,38,38,30,32 | -0.1 (1.18) | -0.3 (0.82) | -0.5 (1.18) | -0.2 (1.02) | 0.1 (1.23) | -0.4 (0.94)
  Direct bilirubin; Week 8; n= 35,37,34, 38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Direct bilirubin; Week 8; n= 35,37,34, 38,29,28 | 0.1 (1.41) | -0.2 (0.99) | -0.4 (1.08) | -0.2 (1.26) | 0.1 (1.36) | -0.5 (1.17)
  Direct bilirubin; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Direct bilirubin; Week 12; n= 36,37,32,35,28,28 | 0.3 (1.19) | 0.0 (1.15) | -0.4 (0.94) | -0.2 (1.17) | 0.0 (1.33) | -0.1 (1.21)
  Direct bilirubin; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Direct bilirubin; Week 14; n= 33,35,32,34,31,29 | -0.1 (1.17) | -0.2 (1.32) | 0.1 (1.19) | -0.2 (1.07) | 0.0 (1.26) | -0.3 (1.58)
  Direct bilirubin; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Direct bilirubin; EW; n= 3,3,7,3,11,11 | 0.0 (2.00) | -0.7 (1.15) | -0.6 (0.98) | -0.7 (1.15) | -0.5 (1.81) | 0.0 (1.26)
  Total bilirubin; Week 2; n=38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Total bilirubin; Week 2; n=38,39,38,39,33,32 | -1.1 (3.21) | -0.8 (3.23) | -2.2 (3.37) | -0.6 (2.64) | -0.4 (5.49) | -0.1 (2.80)
  Total bilirubin; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Total bilirubin; Week 4; n= 38,39,38,38,30,32 | -1.2 (3.18) | -0.8 (2.54) | -1.5 (3.11) | -1.4 (3.15) | 0.3 (4.27) | 0.0 (2.16)
  Total bilirubin; Week 8; n= 35,37,34, 38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Total bilirubin; Week 8; n= 35,37,34, 38,29,28 | 0.0 (4.97) | -0.3 (2.93) | -1.8 (3.24) | -0.8 (4.50) | -0.1 (5.06) | -1.1 (2.14)
  Total bilirubin; Weel 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Total bilirubin; Weel 12; n= 36,37,32,35,28,28 | 0.5 (4.15) | 0.1 (2.26) | -1.9 (2.56) | -0.9 (3.30) | 0.6 (4.42) | -0.1 (3.17)
  Total bilirubin; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Total bilirubin; Week 14; n= 33,35,32,34,31,29 | -0.1 (2.81) | -0.4 (3.90) | 0.0 (4.10) | -0.6 (3.43) | 0.1 (3.92) | -0.4 (4.19)
  Total bilirubin; EW; n = 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Total bilirubin; EW; n = 3,3,7,3,11,11 | -1.3 (5.77) | -2.0 (2.00) | -0.9 (3.44) | -0.7 (1.15) | 0.5 (4.82) | -0.4 (4.27)
  Creatinine; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Creatinine; Week 2; n= 38,39,38,39,33,32 | -3.00 (10.771) | -3.65 (6.186) | -3.46 (7.165) | -0.84 (7.294) | -1.56 (10.461) | 0.11 (8.059)
  Creatinine; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Creatinine; Week 4; n= 38,39,38,38,30,32 | -0.04 (11.471) | -3.30 (6.974) | -1.14 (7.897) | 0.51 (8.990) | -1.19 (10.945) | 3.70 (14.019)
  Creatinine; Week 8; n= 35,37,34, 38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Creatinine; Week 8; n= 35,37,34, 38,29,28 | -2.03 (12.571) | -1.70 (8.249) | -0.29 (8.357) | -0.04 (8.114) | -0.58 (11.799) | -0.51 (7.530)
  Creatinine; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Creatinine; Week 12; n= 36,37,32,35,28,28 | -1.84 (11.918) | -1.41 (9.573) | 0.16 (5.886) | 1.03 (7.618) | -0.70 (10.789) | 1.58 (6.241)
  Creatinine; Week 14; n= 33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Creatinine; Week 14; n= 33,35,32,34,31,29 | 2.04 (10.306) | -1.48 (9.986) | 2.77 (7.351) | 3.17 (7.990) | -0.05 (7.859) | 1.52 (5.860)
  Creatinine; EW; n=3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Creatinine; EW; n=3,3,7,3,11,11 | 1.20 (2.651) | -5.33 (2.650) | -8.19 (9.071) | -4.13 (8.251) | -1.35 (8.386) | 0.09 (11.172)
  Urate; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Urate; Week 2; n= 38,39,38,39,33,32 | -26.1 (74.09) | -7.9 (41.56) | -14.5 (43.91) | 7.9 (49.96) | 0.0 (50.19) | 2.5 (38.44)
  Urate; Week 4; n=38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Urate; Week 4; n=38,39,38,38,30,32 | -18.7 (58.92) | -8.7 (39.21) | -2.9 (52.96) | 3.9 (59.84) | -2.7 (62.69) | 24.1 (62.21)
  Urate; Week 8; n=35,37,34, 38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Urate; Week 8; n=35,37,34, 38,29,28 | -20.0 (60.44) | -0.5 (52.54) | -7.9 (51.63) | -5.5 (59.76) | 12.8 (44.07) | 12.9 (59.25)
  Urate; Week 12; n=36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Urate; Week 12; n=36,37,32,35,28,28 | -20.8 (70.48) | -5.1 (93.20) | -14.7 (46.97) | 2.6 (60.89) | 6.8 (51.43) | 5.0 (46.79)
  Urate; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Urate; Week 14; n=33,35,32,34,31,29 | -10.9 (58.44) | -5.4 (46.86) | 3.8 (48.64) | 15.9 (61.50) | 5.2 (56.32) | 17.2 (43.33)
  Urate; EW; n=3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Urate; EW; n=3,3,7,3,11,11 | -6.7 (20.82) | -16.7 (15.28) | -22.9 (39.46) | -16.7 (85.05) | 0.9 (42.30) | 8.2 (43.55)

23. Secondary Outcome: Change From Baseline in Calcium, Chloride, Carbon Dioxide (CO2), Glucose, Potassium, Sodium, Blood Urea Nitrogen (BUN)
Description: Blood samples were collected to evaluate change from Baseline in calcium, chloride, CO2, glucose, potassium, sodium and BUN values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Millimoles per liter (mmol/L)
  Calcium; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Calcium; Week 2; n= 38,39,38,39,33,32 | -0.042 (0.0941) | -0.037 (0.0918) | -0.067 (0.0970) | -0.022 (0.0822) | -0.024 (0.1346) | -0.027 (0.0758)
  Calcium; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Calcium; Week 4; n= 38,39,38,38,30,32 | -0.037 (0.1076) | -0.014 (0.0899) | -0.050 (0.0873) | -0.028 (0.0840) | -0.031 (0.0952) | -0.031 (0.0900)
  Calcium; Week 8; n=35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Calcium; Week 8; n=35,37,34,38,29,28 | -0.053 (0.0939) | -0.024 (0.0973) | -0.063 (0.0800) | -0.025 (0.0754) | -0.035 (0.0989) | -0.038 (0.0788)
  Calcium; Week 12; n=36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Calcium; Week 12; n=36,37,32,35,28,28 | -0.022 (0.0928) | -0.028 (0.0861) | -0.061 (0.0934) | -0.029 (0.0911) | -0.026 (0.1112) | -0.004 (0.0596)
  Calcium; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Calcium; Week 14; n=33,35,32,34,31,29 | -0.022 (0.0793) | -0.019 (0.0787) | -0.037 (0.0964) | -0.019 (0.0868) | -0.028 (0.0897) | -0.024 (0.0668)
  Calcium; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Calcium; EW; n= 3,3,7,3,11,11 | -0.073 (0.1102) | -0.053 (0.1405) | -0.003 (0.1122) | -0.047 (0.0503) | -0.025 (0.1092) | -0.038 (0.0914)
  Chloride; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Chloride; Week 2; n= 38,39,38,39,33,32 | 0.5 (2.68) | 0.9 (2.32) | 0.2 (2.68) | 0.6 (2.22) | -0.5 (2.49) | 0.4 (2.27)
  Chloride; Week 4; n=38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Chloride; Week 4; n=38,39,38,38,30,32 | 0.5 (2.54) | 0.1 (2.31) | 0.5 (2.05) | 0.3 (2.26) | -0.4 (2.01) | 0.5 (2.38)
  Chloride; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Chloride; Week 8; n= 35,37,34,38,29,28 | 1.0 (2.32) | 0.5 (1.99) | 0.5 (2.27) | -0.3 (2.45) | -0.4 (2.21) | 0.5 (2.86)
  Chloride; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Chloride; Week 12; n= 36,37,32,35,28,28 | 0.1 (2.57) | 0.7 (2.31) | 0.3 (1.85) | 0.5 (2.44) | -0.4 (1.83) | -0.1 (2.76)
  Chloride; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Chloride; Week 14; n=33,35,32,34,31,29 | 0.9 (2.34) | 0.4 (1.82) | 0.1 (2.87) | -0.1 (2.40) | -0.3 (2.32) | 0.6 (2.64)
  Chloride; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Chloride; EW; n= 3,3,7,3,11,11 | -1.0 (1.00) | 1.3 (1.53) | 0.3 (1.98) | 1.0 (2.00) | 0.1 (1.70) | 0.6 (2.66)
  CO2; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  CO2; Week 2; n= 38,39,38,39,33,32 | -1.8 (2.04) | -0.8 (2.52) | -1.2 (2.30) | -0.4 (2.47) | -0.9 (2.39) | -1.0 (2.15)
  CO2; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  CO2; Week 4; n= 38,39,38,38,30,32 | -1.4 (1.98) | -0.8 (3.07) | -1.3 (2.14) | -0.7 (2.22) | -0.5 (2.71) | -1.0 (2.06)
  CO2; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  CO2; Week 8; n= 35,37,34,38,29,28 | -1.9 (2.34) | -1.1 (3.35) | -1.1 (2.21) | -0.7 (2.60) | -0.8 (2.43) | -1.8 (2.65)
  CO2; Week 12; n=36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  CO2; Week 12; n=36,37,32,35,28,28 | -1.1 (2.12) | -1.0 (3.20) | -1.1 (2.45) | -0.7 (2.10) | -0.5 (2.49) | -1.1 (2.07)
  CO2; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  CO2; Week 14; n=33,35,32,34,31,29 | -1.1 (2.23) | -0.8 (3.09) | -1.3 (2.59) | -0.6 (3.13) | -0.9 (2.29) | -1.3 (1.86)
  CO2; EW; n=3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  CO2; EW; n=3,3,7,3,11,11 | 0.0 (1.00) | -0.3 (2.08) | -1.9 (3.18) | 0.3 (1.53) | 0.0 (2.19) | -0.4 (1.80)
  Glucose; Week 2; n=38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Glucose; Week 2; n=38,39,38,39,33,32 | 0.55 (1.710) | 0.65 (1.384) | 0.13 (1.084) | 0.37 (1.431) | 0.46 (0.687) | -0.10 (3.059)
  Glucose; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Glucose; Week 4; n= 38,39,38,38,30,32 | 0.53 (1.334) | 0.25 (1.101) | 0.02 (1.089) | 0.64 (1.209) | 0.38 (1.154) | -0.00 (3.164)
  Glucose; Week 8; n=35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Glucose; Week 8; n=35,37,34,38,29,28 | 0.40 (1.450) | 0.42 (1.253) | 0.01 (0.942) | 0.51 (1.106) | 0.44 (1.048) | -0.34 (3.256)
  Glucose; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Glucose; Week 12; n= 36,37,32,35,28,28 | 0.22 (1.664) | 0.16 (0.990) | 0.01 (1.097) | 0.36 (1.077) | 0.50 (1.028) | -0.49 (3.240)
  Glucose; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Glucose; Week 14; n=33,35,32,34,31,29 | 0.29 (1.091) | 0.47 (1.275) | -0.14 (1.465) | 0.14 (1.482) | 0.12 (0.868) | -0.52 (3.871)
  Glucose; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Glucose; EW; n= 3,3,7,3,11,11 | -0.30 (0.557) | -0.70 (0.889) | 0.67 (1.154) | -0.10 (2.007) | 0.32 (0.873) | 0.11 (0.997)
  Potassium; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Potassium; Week 2; n= 38,39,38,39,33,32 | -0.06 (0.318) | 0.04 (0.360) | 0.04 (0.359) | 0.03 (0.381) | 0.08 (0.371) | 0.03 (0.339)
  Potassium; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Potassium; Week 4; n= 38,39,38,38,30,32 | -0.02 (0.359) | 0.09 (0.446) | 0.19 (0.740) | 0.01 (0.337) | 0.04 (0.254) | 0.01 (0.428)
  Potassium; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Potassium; Week 8; n= 35,37,34,38,29,28 | 0.05 (0.389) | 0.09 (0.303) | 0.19 (0.765) | 0.03 (0.316) | 0.04 (0.344) | -0.06 (0.370)
  Potassium; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Potassium; Week 12; n= 36,37,32,35,28,28 | 0.04 (0.371) | 0.13 (0.335) | -0.01 (0.449) | -0.01 (0.339) | 0.06 (0.398) | 0.01 (0.403)
  Potassium; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Potassium; Week 14; n=33,35,32,34,31,29 | 0.09 (0.309) | 0.13 (0.422) | 0.09 (0.570) | 0.03 (0.349) | 0.14 (0.503) | -0.00 (0.348)
  Potassium; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Potassium; EW; n= 3,3,7,3,11,11 | -0.20 (0.100) | -0.13 (0.208) | 0.10 (0.252) | -0.37 (0.058) | -0.02 (0.236) | -0.00 (0.366)
  Sodium; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Sodium; Week 2; n= 38,39,38,39,33,32 | -0.5 (2.19) | 0.1 (2.17) | -0.1 (2.33) | -0.3 (2.19) | -0.4 (1.90) | -0.2 (1.60)
  Sodium; Week 4; n= 38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Sodium; Week 4; n= 38,39,38,38,30,32 | -0.1 (2.16) | -0.5 (1.94) | -0.2 (1.78) | -0.9 (1.83) | -0.3 (2.14) | -0.1 (1.65)
  Sodium; Week 8; n=35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Sodium; Week 8; n=35,37,34,38,29,28 | -0.3 (2.19) | -0.2 (2.75) | -0.2 (2.21) | -0.7 (1.94) | -0.6 (1.84) | -0.0 (2.50)
  Sodium; Week 12; n=36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Sodium; Week 12; n=36,37,32,35,28,28 | -0.4 (2.11) | -0.4 (2.30) | -0.1 (2.06) | -0.8 (2.02) | -0.8 (2.14) | -0.3 (2.14)
  Sodium; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Sodium; Week 14; n=33,35,32,34,31,29 | 0.2 (1.97) | -0.6 (1.75) | -0.2 (2.34) | -1.0 (2.00) | -0.7 (2.22) | -0.1 (1.93)
  Sodium; EW; n=3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Sodium; EW; n=3,3,7,3,11,11 | -1.3 (1.15) | -1.3 (2.08) | -2.0 (1.00) | -0.3 (0.58) | 0.1 (1.58) | 0.5 (2.34)
  BUN; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  BUN; Week 2; n= 38,39,38,39,33,32 | -0.38 (1.205) | -0.33 (1.078) | 0.03 (1.026) | 0.10 (1.001) | 0.29 (1.256) | -0.19 (1.098)
  BUN; Week 4; n=38,39,38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  BUN; Week 4; n=38,39,38,38,30,32 | -0.38 (1.142) | -0.21 (1.276) | 0.00 (1.202) | -0.08 (1.094) | 0.10 (1.367) | -0.11 (1.091)
  BUN; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  BUN; Week 8; n= 35,37,34,38,29,28 | -0.27 (1.251) | 0.08 (1.199) | -0.03 (0.807) | -0.18 (1.099) | 0.17 (1.159) | 0.02 (1.572)
  BUN; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  BUN; Week 12; n= 36,37,32,35,28,28 | -0.38 (1.250) | -0.09 (1.767) | -0.05 (1.080) | 0.07 (1.030) | 0.23 (1.384) | 0.07 (1.614)
  BUN; Week 14; n=33,35,32,34,31,29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  BUN; Week 14; n=33,35,32,34,31,29 | 0.02 (1.361) | 0.21 (1.540) | 0.19 (1.148) | 0.15 (1.209) | 0.02 (1.268) | 0.19 (1.429)
  BUN; EW; n= 3,3,7,3,11,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  BUN; EW; n= 3,3,7,3,11,11 | -0.33 (0.577) | -0.50 (1.000) | -0.36 (1.144) | -1.00 (0.866) | 0.50 (0.775) | -0.23 (1.915)

24. Secondary Outcome: Number of Participants With Chemistry Data of Potential Clinical Importance
Description: Blood samples were collected from participants for evaluation of clinical chemistry parameters by Potential Clinical Importance Criteria from Baseline to Week 14, EW and any visit post-screen. The vital signs included alk.phosph., ALT, AST, bilirubin, calcium, CO2, creatinine, glucose and potassium. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  Alk.Phosph;Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 0
  Alk.Phosph; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Alk.Phosph; Week 2; n= 38,39,38,39,33,32 | 1 | 0 | 0 | 0 | 0 | 0
  Alk.Phosph.; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Alk.Phosph.; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 0
  Alk.Phosph.; Week 8; n= 35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Alk.Phosph.; Week 8; n= 35, 37, 34, 38, 29, 28 | 1 | 0 | 0 | 0 | 0 | 0
  Alk.Phosph.; Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Alk.Phosph.; Week 12; n= 36, 37, 32, 35, 28, 28 | 1 | 0 | 0 | 0 | 0 | 0
  Alk.Phosph.; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Alk.Phosph.; Week 14; n= 33, 35, 32, 34, 31, 29 | 0 | 0 | 0 | 0 | 0 | 0
  Alk.Phosph.; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Alk.Phosph.; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 0 | 0 | 0
  Alk. Phosph.; post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Alk. Phosph.; post-screen; n= 40, 40,40,39,39,40 | 1 | 0 | 0 | 0 | 0 | 0
  ALT; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 0
  ALT; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  ALT; Week 2; n= 38,39,38,39,33,32 | 1 | 0 | 1 | 0 | 0 | 0
  ALT; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  ALT; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 0
  ALT; Week 8; n=35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  ALT; Week 8; n=35, 37, 34, 38, 29, 28 | 1 | 0 | 0 | 0 | 0 | 0
  ALT; Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  ALT; Week 12; n= 36, 37, 32, 35, 28, 28 | 1 | 0 | 0 | 0 | 0 | 0
  ALT; Week 14; n=33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  ALT; Week 14; n=33, 35, 32, 34, 31, 29 | 1 | 0 | 0 | 0 | 0 | 0
  ALT; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  ALT; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 1 | 0 | 0 | 0
  ALT; post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  ALT; post-screen; n= 40, 40,40,39,39,40 | 2 | 0 | 2 | 0 | 0 | 0
  AST; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 0
  AST; Week 2; n=38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  AST; Week 2; n=38,39,38,39,33,32 | 0 | 0 | 0 | 0 | 0 | 0
  AST; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  AST; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 0
  AST; Week 8; n= 35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  AST; Week 8; n= 35, 37, 34, 38, 29, 28 | 2 | 0 | 0 | 0 | 0 | 0
  AST; Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  AST; Week 12; n= 36, 37, 32, 35, 28, 28 | 0 | 0 | 0 | 0 | 0 | 0
  AST; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  AST; Week 14; n= 33, 35, 32, 34, 31, 29 | 2 | 0 | 0 | 0 | 0 | 0
  AST; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  AST; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 0 | 0 | 0
  AST; Post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  AST; Post-screen; n= 40, 40,40,39,39,40 | 4 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 1 | 0
  Bilirubin; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Bilirubin; Week 2; n= 38,39,38,39,33,32 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Bilirubin; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 1
  Bilirubin; Week 8; n= 35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Bilirubin; Week 8; n= 35, 37, 34, 38, 29, 28 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Week 12; n=36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Bilirubin; Week 12; n=36, 37, 32, 35, 28, 28 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Bilirubin; Week 14; n= 33, 35, 32, 34, 31, 29 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Bilirubin; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin; post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Bilirubin; post-screen; n= 40, 40,40,39,39,40 | 0 | 0 | 1 | 0 | 0 | 1
  Calcium; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Week 2; n=38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Calcium; Week 2; n=38,39,38,39,33,32 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Calcium; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Week 8; n= 35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Calcium; Week 8; n= 35, 37, 34, 38, 29, 28 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Calcium; Week 12; n= 36, 37, 32, 35, 28, 28 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Calcium; Week 14; n= 33, 35, 32, 34, 31, 29 | 0 | 0 | 1 | 0 | 0 | 0
  Calcium; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Calcium; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Calcium; post-screen; n= 40, 40,40,39,39,40 | 0 | 0 | 1 | 0 | 0 | 0
  CO2; Baseline; n= 40,41,43,41,42,40 | 0 | 1 | 0 | 1 | 0 | 0
  CO2; Week 2; n=38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  CO2; Week 2; n=38,39,38,39,33,32 | 1 | 1 | 1 | 0 | 0 | 1
  CO2; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  CO2; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 1 | 0 | 0 | 0
  CO2; Week 8; n= 35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  CO2; Week 8; n= 35, 37, 34, 38, 29, 28 | 1 | 1 | 0 | 1 | 0 | 2
  CO2; Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  CO2; Week 12; n= 36, 37, 32, 35, 28, 28 | 0 | 0 | 0 | 1 | 0 | 0
  CO2; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  CO2; Week 14; n= 33, 35, 32, 34, 31, 29 | 1 | 0 | 2 | 1 | 1 | 0
  CO2; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  CO2; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 0 | 0 | 0
  CO2; Post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  CO2; Post-screen; n= 40, 40,40,39,39,40 | 3 | 2 | 4 | 3 | 1 | 3
  Creatinine; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Creatinine; Week 2; n= 38,39,38,39,33,32 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Creatinine; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine; Week 8; n= 35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Creatinine; Week 8; n= 35, 37, 34, 38, 29, 28 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Creatinine; Week 12; n= 36, 37, 32, 35, 28, 28 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Creatinine; Week 14; n= 33, 35, 32, 34, 31, 29 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Creatinine; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Creatinine; post-screen; n= 40, 40,40,39,39,40 | 0 | 0 | 0 | 0 | 0 | 1
  Glucose; Baseline; n= 40,41,43,41,42,40 | 0 | 1 | 2 | 2 | 1 | 2
  Glucose; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Glucose; Week 2; n= 38,39,38,39,33,32 | 2 | 2 | 0 | 3 | 0 | 2
  Glucose; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Glucose; Week 4; n= 38,39, 38,38,30,32 | 1 | 1 | 0 | 2 | 0 | 3
  Glucose; Week 8; n=35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Glucose; Week 8; n=35, 37, 34, 38, 29, 28 | 1 | 2 | 1 | 2 | 0 | 2
  Glucose; Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Glucose; Week 12; n= 36, 37, 32, 35, 28, 28 | 2 | 1 | 1 | 1 | 0 | 2
  Glucose; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Glucose; Week 14; n= 33, 35, 32, 34, 31, 29 | 0 | 2 | 0 | 3 | 0 | 1
  Glucose; EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Glucose; EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 1 | 0 | 0
  Glucose; post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Glucose; post-screen; n= 40, 40,40,39,39,40 | 4 | 4 | 1 | 6 | 0 | 5
  Potassium; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium; Week 2; n= 38,39,38,39,33,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 33 | 32
  Potassium; Week 2; n= 38,39,38,39,33,32 | 0 | 0 | 0 | 1 | 1 | 0
  Potassium; Week 4; n= 38,39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Potassium; Week 4; n= 38,39, 38,38,30,32 | 0 | 0 | 2 | 0 | 0 | 0
  Potassium; Week 8; n= 35, 37, 34, 38, 29, 28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  Potassium; Week 8; n= 35, 37, 34, 38, 29, 28 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium; n= Week 12; n= 36, 37, 32, 35, 28, 28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Potassium; n= Week 12; n= 36, 37, 32, 35, 28, 28 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium; Week 14; n= 33, 35, 32, 34, 31, 29: number analyzed (Participants) | 33 | 35 | 32 | 34 | 31 | 29
  Potassium; Week 14; n= 33, 35, 32, 34, 31, 29 | 0 | 0 | 1 | 0 | 1 | 0
  Potassium;EW; n= 3, 3, 7, 3, 11, 11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 11 | 11
  Potassium;EW; n= 3, 3, 7, 3, 11, 11 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium; post-screen; n= 40, 40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Potassium; post-screen; n= 40, 40,40,39,39,40 | 0 | 0 | 2 | 1 | 1 | 0

25. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet, Leukocytes Count
Description: Blood samples were collected to evaluate change from Baseline in basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelet and leukocytes and values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter (GI/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Giga cells per liter (GI/L)
  Basophils; Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Basophils; Week 2; n= 37,38,38,37,33,31 | -0.006 (0.0177) | -0.001 (0.0205) | -0.000 (0.0201) | -0.002 (0.0175) | -0.004 (0.0166) | 0.000 (0.0176)
  Basophils; Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Basophils; Week 4; n= 38,38,38,37,30,31 | -0.002 (0.0195) | 0.000 (0.0201) | 0.005 (0.0241) | -0.000 (0.0191) | -0.006 (0.0192) | 0.006 (0.0218)
  Basophils; Week 8; n= 34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Basophils; Week 8; n= 34,36,34,37,29,27 | -0.004 (0.0224) | -0.001 (0.0214) | 0.000 (0.0165) | -0.007 (0.0161) | -0.005 (0.0218) | 0.004 (0.0162)
  Basophils; Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Basophils; Week 12; n= 36,36,32,34,28,27 | 0.001 (0.0166) | 0.002 (0.0191) | 0.005 (0.0244) | 0.003 (0.0343) | 0.003 (0.0348) | 0.010 (0.0236)
  Basophils; Week 14; n= 33,33,32,32,31,27: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 27
  Basophils; Week 14; n= 33,33,32,32,31,27 | -0.001 (0.0160) | -0.000 (0.0190) | 0.003 (0.0202) | -0.003 (0.0226) | 0.008 (0.0312) | -0.001 (0.0188)
  Basophils; EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Basophils; EW; n= 3,3,7,3,10,10 | -0.000 (0.0173) | 0.020 (0.0100) | 0.007 (0.0180) | 0.017 (0.0115) | 0.011 (0.0110) | -0.005 (0.0264)
  Eosinophils; Week 2; n=37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Eosinophils; Week 2; n=37,38,38,37,33,31 | -0.035 (0.2153) | 0.012 (0.1629) | -0.092 (0.2733) | -0.018 (0.2325) | 0.064 (0.4397) | 0.052 (0.1474)
  Eosinophils; Week 4; n=38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Eosinophils; Week 4; n=38,38,38,37,30,31 | -0.075 (0.3146) | -0.049 (0.2401) | -0.119 (0.3926) | -0.034 (0.2143) | 0.063 (0.4729) | 0.057 (0.1644)
  Eosinophils; Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Eosinophils; Week 8; n=34,36,34,37,29,27 | -0.052 (0.3486) | -0.040 (0.1398) | -0.107 (0.3276) | -0.034 (0.2271) | 0.009 (0.1923) | 0.106 (0.2805)
  Eosinophils; Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Eosinophils; Week 12; n= 36,36,32,34,28,27 | -0.083 (0.3212) | -0.026 (0.1811) | -0.120 (0.3025) | -0.063 (0.1751) | -0.028 (0.2176) | 0.033 (0.1606)
  Eosinophils; Week 14; n= 33,33,32,32,31,27: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 27
  Eosinophils; Week 14; n= 33,33,32,32,31,27 | -0.078 (0.3178) | -0.043 (0.2237) | -0.104 (0.2377) | -0.056 (0.1493) | -0.041 (0.2107) | 0.038 (0.1779)
  Eosinophils; EW; n=3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Eosinophils; EW; n=3,3,7,3,10,10 | 0.113 (0.1501) | 0.117 (0.1680) | -0.220 (0.3114) | 0.047 (0.0643) | 0.065 (0.1905) | 0.062 (0.3301)
  Lymphocytes; Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Lymphocytes; Week 2; n= 37,38,38,37,33,31 | 0.035 (0.4672) | 0.076 (0.5239) | 0.123 (0.5263) | 0.064 (0.3510) | 0.030 (0.4724) | 0.018 (0.4654)
  Lymphocytes; Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Lymphocytes; Week 4; n= 38,38,38,37,30,31 | 0.054 (0.5264) | 0.217 (0.5292) | 0.083 (0.5894) | 0.021 (0.4099) | -0.078 (0.4874) | 0.151 (0.5349)
  Lymphocytes; Week 8; n= 34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Lymphocytes; Week 8; n= 34,36,34,37,29,27 | 0.100 (0.3953) | 0.165 (0.6213) | 0.012 (0.4463) | -0.031 (0.3914) | -0.018 (0.5285) | 0.166 (0.4024)
  Lymphocytes; Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Lymphocytes; Week 12; n= 36,36,32,34,28,27 | 0.045 (0.4806) | 0.232 (0.6258) | 0.061 (0.5758) | 0.072 (0.4836) | -0.034 (0.5779) | 0.116 (0.3819)
  Lymphocytes; Week 14; n= 33,33,32,32,31,27: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 27
  Lymphocytes; Week 14; n= 33,33,32,32,31,27 | 0.030 (0.4869) | 0.146 (0.5891) | -0.093 (0.6048) | 0.195 (0.5632) | -0.035 (0.5757) | 0.184 (0.3451)
  Lymphocytes; EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Lymphocytes; EW; n= 3,3,7,3,10,10 | -0.317 (0.5315) | 0.040 (0.0954) | -0.136 (0.4644) | 0.450 (0.0755) | -0.021 (0.4694) | -0.225 (0.4165)
  Monocytes; Week 2; n=37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Monocytes; Week 2; n=37,38,38,37,33,31 | -0.028 (0.1465) | -0.025 (0.1271) | 0.013 (0.1659) | 0.008 (0.0965) | -0.028 (0.1415) | 0.019 (0.1948)
  Monocytes; Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Monocytes; Week 4; n= 38,38,38,37,30,31 | -0.004 (0.1769) | -0.023 (0.1230) | -0.059 (0.1648) | 0.006 (0.1151) | -0.047 (0.1611) | 0.010 (0.1419)
  Monocytes; Week 8; n= 34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Monocytes; Week 8; n= 34,36,34,37,29,27 | -0.071 (0.1443) | -0.041 (0.1224) | -0.032 (0.1355) | -0.012 (0.1359) | -0.066 (0.1465) | -0.001 (0.1171)
  Monocytes; Week 12; n=36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Monocytes; Week 12; n=36,36,32,34,28,27 | -0.061 (0.1653) | -0.022 (0.1219) | -0.042 (0.1539) | -0.019 (0.1434) | -0.078 (0.1736) | 0.007 (0.1801)
  Monocytes; Week 14; n=33,33,32,32,31,27: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 27
  Monocytes; Week 14; n=33,33,32,32,31,27 | -0.026 (0.1532) | 0.027 (0.1427) | -0.016 (0.1446) | 0.015 (0.1666) | -0.093 (0.1497) | 0.035 (0.1821)
  Monocytes; EW; n=3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Monocytes; EW; n=3,3,7,3,10,10 | -0.127 (0.0924) | 0.007 (0.0850) | 0.030 (0.1133) | 0.040 (0.0608) | -0.018 (0.0966) | -0.159 (0.1672)
  Neutrophils; Week 2; n=37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Neutrophils; Week 2; n=37,38,38,37,33,31 | 0.480 (1.7953) | 0.152 (1.0058) | 0.067 (1.7035) | -0.088 (1.4680) | -0.097 (1.8249) | -0.258 (1.2803)
  Neutrophils; Week 4; n=38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Neutrophils; Week 4; n=38,38,38,37,30,31 | 0.487 (2.0425) | 0.253 (1.1437) | -0.058 (1.7028) | 0.035 (1.3063) | -0.141 (2.1024) | 0.100 (1.4283)
  Neutrophils; Week 8; n= 34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Neutrophils; Week 8; n= 34,36,34,37,29,27 | 0.009 (1.4215) | -0.203 (1.0365) | -0.083 (1.4454) | 0.550 (1.5918) | -0.432 (1.5971) | 0.214 (1.1894)
  Neutrophils; Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Neutrophils; Week 12; n= 36,36,32,34,28,27 | 0.127 (1.3363) | -0.009 (1.1315) | 0.049 (1.4294) | 0.237 (1.1459) | -0.348 (1.5514) | 0.328 (1.6786)
  Neutrophils; Week 14; n=33,33,32,32,31,27: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 27
  Neutrophils; Week 14; n=33,33,32,32,31,27 | 0.090 (1.2037) | 0.164 (1.2465) | -0.368 (1.0224) | -0.058 (1.5202) | -0.155 (1.9840) | -0.013 (1.4826)
  Neutrophils; EW; n=3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Neutrophils; EW; n=3,3,7,3,10,10 | -0.420 (0.9924) | 0.047 (0.7478) | 0.797 (2.1506) | 0.630 (1.0741) | -0.331 (1.2306) | 0.158 (1.8160)
  Platelet; Week 2; n=37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Platelet; Week 2; n=37,38,38,37,33,31 | -15.4 (44.06) | -18.7 (36.48) | -25.9 (43.03) | -20.2 (30.63) | -0.5 (31.18) | 6.9 (31.60)
  Platelet; Week 4; n=38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Platelet; Week 4; n=38,38,38,37,30,31 | -12.4 (36.57) | -19.7 (36.44) | -25.2 (35.75) | -7.7 (38.40) | -2.4 (30.48) | 12.7 (29.38)
  Platelet; Week 8; n= 34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Platelet; Week 8; n= 34,36,34,37,29,27 | -6.2 (34.81) | -9.1 (51.69) | -22.1 (37.57) | -11.5 (44.80) | 1.4 (37.70) | 8.8 (39.83)
  Platelet; Week 12; n=36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Platelet; Week 12; n=36,36,32,34,28,27 | -7.5 (37.94) | -5.4 (30.15) | -23.6 (38.11) | -18.9 (38.67) | -4.6 (35.71) | -6.8 (24.06)
  Platelet; Week 14; n=33,33,32,32,31,27: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 27
  Platelet; Week 14; n=33,33,32,32,31,27 | 3.5 (40.84) | -9.0 (38.20) | -19.9 (44.95) | -8.2 (47.60) | 5.1 (31.34) | 6.5 (51.77)
  Platelet; EW; n=3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Platelet; EW; n=3,3,7,3,10,10 | -85.0 (11.00) | 12.7 (56.01) | -19.7 (25.77) | 11.7 (18.56) | 8.4 (24.56) | 11.3 (59.83)
  Leukocytes; Week 2; n=37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Leukocytes; Week 2; n=37,38,38,37,33,31 | 0.45 (1.749) | 0.21 (1.085) | 0.10 (1.668) | -0.02 (1.585) | -0.05 (1.972) | -0.16 (1.624)
  Leukocytes; Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Leukocytes; Week 4; n= 38,38,38,37,30,31 | 0.46 (1.913) | 0.40 (1.232) | -0.15 (1.807) | 0.03 (1.517) | -0.21 (2.221) | 0.34 (1.694)
  Leukocytes; Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Leukocytes; Week 8; n=34,36,34,37,29,27 | 0.03 (1.466) | -0.12 (1.257) | -0.21 (1.567) | 0.47 (1.469) | -0.52 (1.721) | 0.49 (1.113)
  Leukocytes; Week 12; n=36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Leukocytes; Week 12; n=36,36,32,34,28,27 | 0.03 (1.488) | 0.18 (1.249) | -0.05 (1.371) | 0.23 (1.248) | -0.49 (1.456) | 0.49 (1.776)
  Leukocytes; Week 14; n=33,33,32,32,31,27: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 27
  Leukocytes; Week 14; n=33,33,32,32,31,27 | 0.02 (1.234) | 0.30 (1.200) | -0.57 (1.142) | 0.10 (1.705) | -0.32 (2.121) | 0.23 (1.498)
  Leukocytes; EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Leukocytes; EW; n= 3,3,7,3,10,10 | -0.73 (0.666) | 0.23 (1.115) | 0.47 (2.394) | 1.20 (1.127) | -0.29 (1.454) | -0.16 (2.151)

26. Secondary Outcome: Change From Baseline in Hematocrit Levels
Description: Blood samples were collected to evaluate change from Baseline in hematocrit and values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Proportion of red blood cells in blood
  Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Week 2; n= 37,38,38,37,33,31 | -0.0054 (0.0276) | -0.0132 (0.0195) | -0.0138 (0.0260) | -0.0116 (0.0246) | -0.0014 (0.0267) | -0.0095 (0.0239)
  Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Week 4; n= 38,38,38,37,30,31 | -0.0107 (0.0315) | -0.0075 (0.0241) | -0.0081 (0.0253) | -0.0075 (0.0233) | -0.0090 (0.0283) | -0.0123 (0.0295)
  Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Week 8; n=34,36,34,37,29,27 | -0.0066 (0.0316) | -0.0148 (0.0225) | -0.0091 (0.0225) | -0.0042 (0.0235) | -0.0011 (0.0264) | -0.0124 (0.0314)
  Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Week 12; n= 36,36,32,34,28,27 | -0.0054 (0.0302) | -0.0129 (0.0222) | -0.0131 (0.0205) | -0.0106 (0.0227) | -0.0052 (0.0312) | -0.0111 (0.0240)
  Week 14; n= 33,33,32,32,31,28: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 28
  Week 14; n= 33,33,32,32,31,28 | -0.0151 (0.0292) | -0.0170 (0.0236) | -0.0132 (0.0193) | -0.0063 (0.0286) | -0.0007 (0.0277) | -0.0117 (0.0292)
  EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  EW; n= 3,3,7,3,10,10 | 0.0037 (0.0123) | -0.0063 (0.0352) | -0.0174 (0.0292) | -0.0117 (0.0133) | 0.0027 (0.0152) | 0.0048 (0.0248)

27. Secondary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Blood samples were collected to evaluate change from Baseline in hemoglobin and MCHC and values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
G/L
  Hemoglobin; Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Hemoglobin; Week 2; n= 37,38,38,37,33,31 | -1.8 (9.02) | -3.8 (5.54) | -4.3 (8.08) | -2.8 (6.78) | -0.9 (8.76) | -3.0 (6.55)
  Hemoglobin; Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Hemoglobin; Week 4; n= 38,38,38,37,30,31 | -3.2 (8.88) | -2.7 (6.42) | -3.5 (7.72) | -2.4 (6.27) | -3.0 (9.17) | -4.1 (9.05)
  Hemoglobin; Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Hemoglobin; Week 8; n=34,36,34,37,29,27 | -2.7 (9.64) | -4.6 (6.43) | -3.7 (6.90) | -1.6 (6.70) | -0.8 (7.59) | -4.6 (9.72)
  Hemoglobin; Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Hemoglobin; Week 12; n= 36,36,32,34,28,27 | -2.3 (9.33) | -4.2 (6.61) | -5.2 (6.77) | -3.1 (5.58) | -2.5 (9.52) | -4.4 (6.63)
  Hemoglobin; Week 14; n= 33,33,32,32,31,28: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 28
  Hemoglobin; Week 14; n= 33,33,32,32,31,28 | -5.5 (9.25) | -3.9 (6.76) | -5.2 (6.73) | -1.8 (8.17) | -0.8 (8.51) | -4.0 (7.93)
  Hemoglobin; EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Hemoglobin; EW; n= 3,3,7,3,10,10 | 0.7 (11.59) | -1.3 (11.59) | -6.0 (8.47) | -2.0 (9.00) | 0.0 (3.77) | -1.1 (5.69)
  MCHC; Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  MCHC; Week 2; n= 37,38,38,37,33,31 | 0.1 (7.47) | 0.9 (7.83) | 0.8 (6.65) | 2.0 (10.23) | -1.4 (8.37) | 8.37 (8.92)
  MCHC; Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  MCHC; Week 4; n= 38,38,38,37,30,31 | 0.9 (8.89) | -0.3 (9.51) | -1.9 (9.53) | 0.2 (9.62) | 0.0 (9.14) | 0.1 (8.17)
  MCHC; Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  MCHC; Week 8; n=34,36,34,37,29,27 | -1.1 (9.28) | 0.4 (11.61) | -1.9 (8.69) | -0.5 (11.02) | -0.5 (10.28) | -1.3 (8.96)
  MCHC; Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  MCHC; Week 12; n= 36,36,32,34,28,27 | -1.0 (10.23) | 0.1 (11.12) | -2.5 (10.95) | 0.9 (10.85) | -1.4 (10.77) | -1.8 (9.95)
  MCHC; Week 14; n= 33,33,32,32,31,28: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 28
  MCHC; Week 14; n= 33,33,32,32,31,28 | -1.2 (11.15) | 3.9 (10.96) | -2.2 (10.24) | 0.7 (10.42) | -1.0 (11.18) | -0.1 (8.59)
  MCHC; EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  MCHC; EW; n= 3,3,7,3,10,10 | -1.7 (20.26) | 1.7 (2.52) | -1.1 (10.64) | 3.3 (12.86) | -2.2 (5.25) | -6.6 (9.09)

28. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH)
Description: Blood samples were collected to evaluate change from Baseline in MCH and values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picogram (Pg)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Picogram (Pg)
  Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Week 2; n= 37,38,38,37,33,31 | 0.05 (0.425) | 0.09 (0.595) | 0.06 (0.408) | 0.19 (0.667) | 0.04 (0.415) | 0.05 (0.490)
  Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Week 4; n= 38,38,38,37,30,31 | 0.09 (0.535) | 0.06 (0.593) | -0.01 (0.519) | 0.15 (0.567) | 0.06 (0.518) | -0.05 (0.528)
  Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Week 8; n=34,36,34,37,29,27 | 0.03 (0.635) | 0.21 (0.747) | -0.06 (0.536) | 0.22 (0.781) | 0.02 (0.599) | -0.07 (0.640)
  Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Week 12; n= 36,36,32,34,28,27 | 0.14 (0.708) | 0.14 (0.790) | 0.10 (0.506) | 0.30 (0.815) | 0.04 (0.588) | 0.06 (0.806)
  Week 14; n= 33,33,32,32,31,28: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 28
  Week 14; n= 33,33,32,32,31,28 | 0.06 (0.900) | 0.55 (0.806) | 0.08 (0.449) | 0.28 (0.612) | 0.06 (0.804) | -0.01 (0.589)
  EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  EW; n= 3,3,7,3,10,10 | 0.57 (1.361) | 0.03 (0.702) | -0.19 (0.596) | 0.63 (0.808) | -0.13 (0.933) | -0.15 (0.542)

29. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV)
Description: Blood samples were collected to evaluate change from Baseline in MCV and values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Femtoliter (fL)
  Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Week 2; n= 37,38,38,37,33,31 | 0.2 (2.02) | -0.2 (1.45) | -0.1 (1.47) | -0.1 (2.37) | 0.5 (1.87) | 0.1 (1.83)
  Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Week 4; n= 38,38,38,37,30,31 | 0.1 (1.75) | 0.2 (2.04) | 0.5 (1.94) | 0.4 (2.80) | 0.1 (1.90) | -0.3 (1.85)
  Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Week 8; n=34,36,34,37,29,27 | 0.5 (2.42) | 0.5 (2.52) | 0.4 (1.78) | 0.7 (2.90) | 0.2 (2.39) | 0.0 (2.01)
  Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Week 12; n= 36,36,32,34,28,27 | 0.8 (2.80) | 0.3 (2.68) | 1.0 (2.62) | 0.6 (3.20) | 0.5 (3.06) | 0.5 (1.99)
  Week 14; n= 33,33,32,32,31,28: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 28
  Week 14; n= 33,33,32,32,31,28 | 0.6 (2.92) | 0.4 (2.54) | 0.9 (2.54) | 0.7 (2.37) | 0.4 (3.19) | -0.1 (2.25)
  EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  EW; n= 3,3,7,3,10,10 | 1.7 (1.53) | -0.7 (2.08) | -0.4 (2.15) | 1.0 (1.00) | -0.1 (2.81) | 1.4 (2.59)

30. Secondary Outcome: Change From Baseline in Erythrocyte Count
Description: Blood samples were collected to evaluate change from Baseline in erythrocytes and values at Baseline throughout the 12 weeks of study treatment and follow up visit 1 at Week 14. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Weeks 2, 4, 8, 12, 14, EW (week up to 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Tetra cells per liter (TI/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Tetra cells per liter (TI/L)
  Week 2; n= 37,38,38,37,33,31: number analyzed (Participants) | 37 | 38 | 38 | 37 | 33 | 31
  Week 2; n= 37,38,38,37,33,31 | -0.06 (0.325) | -0.16 (0.218) | -0.15 (0.287) | -0.12 (0.260) | -0.03 (0.293) | -0.12 (0.241)
  Week 4; n= 38,38,38,37,30,31: number analyzed (Participants) | 38 | 38 | 38 | 37 | 30 | 31
  Week 4; n= 38,38,38,37,30,31 | -0.12 (0.347) | -0.10 (0.256) | -0.13 (0.273) | -0.10 (0.215) | -0.11 (0.317) | -0.13 (0.312)
  Week 8; n=34,36,34,37,29,27: number analyzed (Participants) | 34 | 36 | 34 | 37 | 29 | 27
  Week 8; n=34,36,34,37,29,27 | -0.10 (0.371) | -0.21 (0.227) | -0.12 (0.265) | -0.08 (0.205) | -0.03 (0.268) | -0.14 (0.318)
  Week 12; n= 36,36,32,34,28,27: number analyzed (Participants) | 36 | 36 | 32 | 34 | 28 | 27
  Week 12; n= 36,36,32,34,28,27 | -0.09 (0.345) | -0.18 (0.244) | -0.21 (0.250) | -0.15 (0.191) | -0.09 (0.314) | -0.15 (0.262)
  Week 14; n= 33,33,32,32,31,28: number analyzed (Participants) | 33 | 33 | 32 | 32 | 31 | 28
  Week 14; n= 33,33,32,32,31,28 | -0.20 (0.342) | -0.22 (0.262) | -0.21 (0.229) | -0.10 (0.261) | -0.03 (0.330) | -0.14 (0.312)
  EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  EW; n= 3,3,7,3,10,10 | -0.03 (0.252) | -0.07 (0.321) | -0.19 (0.297) | -0.13 (0.153) | 0.04 (0.246) | -0.03 (0.267)

31. Secondary Outcome: Number of Participants With Hematology Data of Potential Clinical Importance
Description: Blood samples were collected from participants for evaluation of hematology parameters by Potential Clinical Importance Criteria from Baseline to Week 14, EW and any visit post-screen. The vital signs included hematocrit, hemoglobin, lymphocytes, neutrophils, platelet and leukocytes. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline, Week 2, 4, 8, 12, 14, early withdrawal, and post screen (up to Week 16)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  Hematocrit; Baseline; n= 40, 40, 43, 40, 42, 39: number analyzed (Participants) | 40 | 40 | 43 | 40 | 42 | 39
  Hematocrit; Baseline; n= 40, 40, 43, 40, 42, 39 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit; Week 2; n= 37, 39, 38, 38, 33, 31: number analyzed (Participants) | 37 | 39 | 38 | 38 | 33 | 31
  Hematocrit; Week 2; n= 37, 39, 38, 38, 33, 31 | 0 | 0 | 0 | 0 | 1 | 0
  Hematocrit; Week 4; n= 38, 39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Hematocrit; Week 4; n= 38, 39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 1
  Hematocrit; Week 8; n=34,36,34,38,29,28: number analyzed (Participants) | 34 | 36 | 34 | 38 | 29 | 28
  Hematocrit; Week 8; n=34,36,34,38,29,28 | 1 | 0 | 1 | 0 | 1 | 1
  Hematocrit; Week 12; n= 36, 37, 32, 35, 28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Hematocrit; Week 12; n= 36, 37, 32, 35, 28,28 | 1 | 0 | 0 | 0 | 0 | 0
  Hematocrit; Week 14; n= 33,34,32,33,31,29: number analyzed (Participants) | 33 | 34 | 32 | 33 | 31 | 29
  Hematocrit; Week 14; n= 33,34,32,33,31,29 | 1 | 0 | 0 | 0 | 0 | 2
  Hematocrit; EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Hematocrit; EW; n= 3,3,7,3,10,10 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit; post-screen; n= 40,40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Hematocrit; post-screen; n= 40,40,40,39,39,40 | 2 | 0 | 1 | 0 | 1 | 2
  Hemoglobin; Baseline;n= 40, 40, 43, 40, 42, 39: number analyzed (Participants) | 40 | 40 | 43 | 40 | 42 | 39
  Hemoglobin; Baseline;n= 40, 40, 43, 40, 42, 39 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin; Week 2; n= 37, 39, 38, 38, 33, 31: number analyzed (Participants) | 37 | 39 | 38 | 38 | 33 | 31
  Hemoglobin; Week 2; n= 37, 39, 38, 38, 33, 31 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin; Week 4; n= 38, 39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Hemoglobin; Week 4; n= 38, 39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin; Week 8; n= 34,36,34,38,29,28: number analyzed (Participants) | 34 | 36 | 34 | 38 | 29 | 28
  Hemoglobin; Week 8; n= 34,36,34,38,29,28 | 1 | 0 | 0 | 0 | 0 | 1
  Hemoglobin; Week 12; n= 36, 37, 32, 35, 28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Hemoglobin; Week 12; n= 36, 37, 32, 35, 28,28 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin; Week 14; n=33,34,32,33,31,29: number analyzed (Participants) | 33 | 34 | 32 | 33 | 31 | 29
  Hemoglobin; Week 14; n=33,34,32,33,31,29 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin; EW; n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Hemoglobin; EW; n= 3,3,7,3,10,10 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin; post-screen; n= 40,40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Hemoglobin; post-screen; n= 40,40,40,39,39,40 | 1 | 0 | 0 | 0 | 0 | 1
  Lymphocytes;Baseline; n= 40, 40, 43, 40, 42, 39: number analyzed (Participants) | 40 | 40 | 43 | 40 | 42 | 39
  Lymphocytes;Baseline; n= 40, 40, 43, 40, 42, 39 | 0 | 1 | 1 | 0 | 0 | 1
  Lymphocytes; Week 2; n= 37, 39, 38, 38, 33, 31: number analyzed (Participants) | 37 | 39 | 38 | 38 | 33 | 31
  Lymphocytes; Week 2; n= 37, 39, 38, 38, 33, 31 | 0 | 1 | 0 | 0 | 0 | 0
  Lymhocytes; Week 4; n= 38, 39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Lymhocytes; Week 4; n= 38, 39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes; Week 8; n= 34,36,34,38,29,28: number analyzed (Participants) | 34 | 36 | 34 | 38 | 29 | 28
  Lymphocytes; Week 8; n= 34,36,34,38,29,28 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes; Week 12; n=36, 37, 32, 35, 28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Lymphocytes; Week 12; n=36, 37, 32, 35, 28,28 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocytes; Week 14; n= 33,34,32,33,31,28: number analyzed (Participants) | 33 | 34 | 32 | 33 | 31 | 28
  Lymphocytes; Week 14; n= 33,34,32,33,31,28 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes; EW;n= 3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Lymphocytes; EW;n= 3,3,7,3,10,10 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes; post-screen; n= 40,40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Lymphocytes; post-screen; n= 40,40,40,39,39,40 | 0 | 1 | 0 | 0 | 1 | 0
  Neutrophils; Baseline; n= 40, 40, 43, 40, 42, 39: number analyzed (Participants) | 40 | 40 | 43 | 40 | 42 | 39
  Neutrophils; Baseline; n= 40, 40, 43, 40, 42, 39 | 2 | 0 | 0 | 0 | 0 | 0
  Neutrophils; Week 2; n= 37, 39, 38, 38, 33, 31: number analyzed (Participants) | 37 | 39 | 38 | 38 | 33 | 31
  Neutrophils; Week 2; n= 37, 39, 38, 38, 33, 31 | 0 | 1 | 0 | 1 | 0 | 0
  Neutrophils; Week 4; n= 38, 39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Neutrophils; Week 4; n= 38, 39, 38,38,30,32 | 4 | 0 | 1 | 0 | 0 | 0
  Neutrophils; Week 8; n= 34,36,34,38,29,28: number analyzed (Participants) | 34 | 36 | 34 | 38 | 29 | 28
  Neutrophils; Week 8; n= 34,36,34,38,29,28 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils; Week 12; n= 36, 37, 32, 35, 28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Neutrophils; Week 12; n= 36, 37, 32, 35, 28,28 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils; Week 14; n=33,34,32,33,31,29: number analyzed (Participants) | 33 | 34 | 32 | 33 | 31 | 29
  Neutrophils; Week 14; n=33,34,32,33,31,29 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils; EW; n=3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Neutrophils; EW; n=3,3,7,3,10,10 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils; post-screen;n= 40,40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Neutrophils; post-screen;n= 40,40,40,39,39,40 | 4 | 2 | 1 | 1 | 0 | 0
  Platelets; Baseline; n= 40, 40, 43, 40, 42, 39: number analyzed (Participants) | 40 | 40 | 43 | 40 | 42 | 39
  Platelets; Baseline; n= 40, 40, 43, 40, 42, 39 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets; Week 2; n= :37,38,38,38,33,31: number analyzed (Participants) | 37 | 38 | 38 | 38 | 33 | 31
  Platelets; Week 2; n= :37,38,38,38,33,31 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets; Week 4; n=37,39, 38,38,30,32: number analyzed (Participants) | 37 | 39 | 38 | 38 | 30 | 32
  Platelets; Week 4; n=37,39, 38,38,30,32 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets; Week 8; n= 34,36,34,38,29,28: number analyzed (Participants) | 34 | 36 | 34 | 38 | 29 | 28
  Platelets; Week 8; n= 34,36,34,38,29,28 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets; Week 12; n= 35,37,32,35,28,28: number analyzed (Participants) | 35 | 37 | 32 | 35 | 28 | 28
  Platelets; Week 12; n= 35,37,32,35,28,28 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets; Week 14; n=33,34,32,33,31,29: number analyzed (Participants) | 33 | 34 | 32 | 33 | 31 | 29
  Platelets; Week 14; n=33,34,32,33,31,29 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets; EW; n=3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Platelets; EW; n=3,3,7,3,10,10 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets; post-screen; n= 40,40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Platelets; post-screen; n= 40,40,40,39,39,40 | 0 | 0 | 0 | 0 | 1 | 1
  Leukocytes; Baseline; n= 40, 40, 43, 40, 42, 39: number analyzed (Participants) | 40 | 40 | 43 | 40 | 42 | 39
  Leukocytes; Baseline; n= 40, 40, 43, 40, 42, 39 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes; Week 2; n=37, 39, 38, 38, 33, 31: number analyzed (Participants) | 37 | 39 | 38 | 38 | 33 | 31
  Leukocytes; Week 2; n=37, 39, 38, 38, 33, 31 | 0 | 1 | 0 | 1 | 0 | 0
  Leukocytes; Week 4; n=38, 39, 38,38,30,32: number analyzed (Participants) | 38 | 39 | 38 | 38 | 30 | 32
  Leukocytes; Week 4; n=38, 39, 38,38,30,32 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes; Week 8; n=34,36,34,38,29,28: number analyzed (Participants) | 34 | 36 | 34 | 38 | 29 | 28
  Leukocytes; Week 8; n=34,36,34,38,29,28 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes; Week 12; n= 36, 37, 32, 35, 28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Leukocytes; Week 12; n= 36, 37, 32, 35, 28,28 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes; Week 14; n=33,34,32,33,31,28: number analyzed (Participants) | 33 | 34 | 32 | 33 | 31 | 28
  Leukocytes; Week 14; n=33,34,32,33,31,28 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes; n= EW; n=3,3,7,3,10,10: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 10
  Leukocytes; n= EW; n=3,3,7,3,10,10 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes; post-screen; n= 40,40,40,39,39,40: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Leukocytes; post-screen; n= 40,40,40,39,39,40 | 0 | 1 | 0 | 1 | 0 | 0

32. Secondary Outcome: Change From Baseline in Total T Lymphocytes (Lympho), B Lympho, Natural Killer (NK) Lymphocytes and Treg (Foxp3) Levels
Description: Blood samples were collected to evaluate change from Baseline in total T lympho, B lympho, T and B NK cells and (Foxp3) values at Baseline throughout the 12 weeks of study treatment. The immunophenotyping parameters included cluster of differentiation (CD)19, CD3, CD3+CD8+, CD3+CD4+, CD16+CD56+, CD3+CD4+CD25+CD127, CD3+CD4+foxP3+CD25+CD127 and T and NK lympho. CD3, CD3+CD8+ and CD3+CD4+ were also evaluated by using treg flow cytometry (cyto). Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week, 4, 8 and 12
Population: Safety population
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
GI/L
  CD19; Week 4; n= 37,38,38,37,29,32: number analyzed (Participants) | 37 | 38 | 38 | 37 | 29 | 32
  CD19; Week 4; n= 37,38,38,37,29,32 | 0.0394 (0.1149) | 0.0407 (0.1229) | 0.0068 (0.1532) | 0.0174 (0.0933) | -0.0217 (0.1410) | 0.0406 (0.1114)
  CD19; Week 8; n=34,37,34,37,28,27: number analyzed (Participants) | 34 | 37 | 34 | 37 | 28 | 27
  CD19; Week 8; n=34,37,34,37,28,27 | 0.0273 (0.0951) | 0.0343 (0.1480) | 0.0122 (0.1154) | -0.0006 (0.1099) | -0.0282 (0.1502) | 0.0367 (0.0966)
  CD19; Week 12; n= 35,37,32,34,27,27: number analyzed (Participants) | 35 | 37 | 32 | 34 | 27 | 27
  CD19; Week 12; n= 35,37,32,34,27,27 | 0.0111 (0.1262) | 0.0647 (0.1440) | 0.0317 (0.1077) | 0.0224 (0.0927) | -0.0439 (0.1350) | 0.0041 (0.1009)
  CD3; Week 4; n= 37,38,38,37,29,32: number analyzed (Participants) | 37 | 38 | 38 | 37 | 29 | 32
  CD3; Week 4; n= 37,38,38,37,29,32 | -0.0050 (0.3830) | 0.0867 (0.3809) | 0.0842 (0.3343) | 0.0108 (0.3364) | -0.0397 (0.4505) | 0.1678 (0.3583)
  CD3; Week 8; n=34,37,34,37,28,27: number analyzed (Participants) | 34 | 37 | 34 | 37 | 28 | 27
  CD3; Week 8; n=34,37,34,37,28,27 | 0.0523 (0.3117) | 0.0581 (0.4496) | 0.0334 (0.3855) | -0.0593 (0.3172) | -0.0350 (0.4403) | 0.1066 (0.3531)
  CD3; Week 12; n= 35,37,32,34,27,27: number analyzed (Participants) | 35 | 37 | 32 | 34 | 27 | 27
  CD3; Week 12; n= 35,37,32,34,27,27 | -0.0045 (0.4254) | 0.1312 (0.4033) | 0.1375 (0.4003) | 0.0071 (0.2729) | -0.1338 (0.5023) | 0.0167 (0.2879)
  CD3 treg flow cyto; Week 4; n= 35,37,36,35,28,28: number analyzed (Participants) | 35 | 37 | 36 | 35 | 28 | 28
  CD3 treg flow cyto; Week 4; n= 35,37,36,35,28,28 | -0.0277 (0.3912) | 0.0643 (0.3988) | 0.0682 (0.2853) | 0.0270 (0.3320) | -0.0688 (0.4764) | 0.1943 (0.3722)
  CD3; treg flow cyto; Week 8; n=31,35,32,36,27,25: number analyzed (Participants) | 31 | 35 | 32 | 36 | 27 | 25
  CD3; treg flow cyto; Week 8; n=31,35,32,36,27,25 | 0.0184 (0.2929) | 0.0745 (0.4592) | -0.0023 (0.3513) | -0.0647 (0.3128) | -0.0626 (0.4679) | 0.1302 (0.3505)
  CD3; treg flow cyto; Week 12; n= 32,36,31,32,25,24: number analyzed (Participants) | 32 | 36 | 31 | 32 | 25 | 24
  CD3; treg flow cyto; Week 12; n= 32,36,31,32,25,24 | -0.0215 (0.4120) | 0.1418 (0.4318) | 0.1171 (0.4070) | -0.0063 (0.2771) | -0.1402 (0.5450) | 0.0028 (0.3101)
  CD3+CD8+; Week 4; n= 37,38,38,37,29,32: number analyzed (Participants) | 37 | 38 | 38 | 37 | 29 | 32
  CD3+CD8+; Week 4; n= 37,38,38,37,29,32 | -0.0272 (0.2077) | 0.0248 (0.1298) | 0.0282 (0.1266) | 0.0147 (0.1194) | -0.0155 (0.1608) | 0.0526 (0.1388)
  CD3+CD8+; Week 8; n= 34,37,34,37,28,27: number analyzed (Participants) | 34 | 37 | 34 | 37 | 28 | 27
  CD3+CD8+; Week 8; n= 34,37,34,37,28,27 | -0.0048 (0.1337) | 0.0011 (0.1561) | 0.0242 (0.1335) | -0.0263 (0.1145) | -0.0315 (0.1677) | 0.0322 (0.1721)
  CD3+CD8+; Week 12;n=35,37,32,34,27,27: number analyzed (Participants) | 35 | 37 | 32 | 34 | 27 | 27
  CD3+CD8+; Week 12;n=35,37,32,34,27,27 | -0.0307 (0.1754) | 0.0270 (0.1392) | 0.0357 (0.1578) | -0.0115 (0.0868) | -0.0853 (0.1818) | -0.0023 (0.1097)
  CD3+CD8+ treg flow cyto;Week 4;n=35,37,36,35,28,28: number analyzed (Participants) | 35 | 37 | 36 | 35 | 28 | 28
  CD3+CD8+ treg flow cyto;Week 4;n=35,37,36,35,28,28 | -0.0392 (0.2124) | 0.0211 (0.1222) | 0.0004 (0.1117) | 0.0038 (0.1112) | -0.0246 (0.1572) | 0.0728 (0.1175)
  CD3+CD8+ treg flow cyto;Week 8;n=31,35,32,36,27,25: number analyzed (Participants) | 31 | 35 | 32 | 36 | 27 | 25
  CD3+CD8+ treg flow cyto;Week 8;n=31,35,32,36,27,25 | 0.0004 (0.1228) | 0.0125 (0.1350) | -0.0008 (0.1214) | -0.0376 (0.1150) | -0.0351 (0.1672) | 0.0484 (0.1417)
  CD3+CD8+treg flow cyto;Week12;n=32,36,31,32,25,24: number analyzed (Participants) | 32 | 36 | 31 | 32 | 25 | 24
  CD3+CD8+treg flow cyto;Week12;n=32,36,31,32,25,24 | -0.0179 (0.1738) | 0.0311 (0.1338) | 0.0151 (0.1490) | -0.0230 (0.0865) | -0.0689 (0.1752) | 0.0120 (0.1064)
  CD3+CD4+; Week 4; n= 37,38,38,37,29,32: number analyzed (Participants) | 37 | 38 | 38 | 37 | 29 | 32
  CD3+CD4+; Week 4; n= 37,38,38,37,29,32 | 0.0080 (0.2066) | 0.0579 (0.2532) | 0.0562 (0.2652) | -0.0030 (0.2342) | -0.0268 (0.2913) | 0.1138 (0.2308)
  CD3+CD4+; Week 8; n=34,37,34,37,28,27: number analyzed (Participants) | 34 | 37 | 34 | 37 | 28 | 27
  CD3+CD4+; Week 8; n=34,37,34,37,28,27 | 0.0282 (0.1739) | 0.0539 (0.2996) | 0.0072 (0.2794) | -0.0287 (0.2054) | -0.0015 (0.2803) | 0.0778 (0.1826)
  CD3+CD4+; Week 12; n= 35,37,32,34,27,27: number analyzed (Participants) | 35 | 37 | 32 | 34 | 27 | 27
  CD3+CD4+; Week 12; n= 35,37,32,34,27,27 | 0.0243 (0.2551) | 0.0957 (0.2713) | 0.1087 (0.2795) | 0.0216 (0.1929) | -0.0465 (0.3338) | 0.0181 (0.1872)
  CD3+CD4+ treg flow cyto;Week 4;n=35,37,36,35,28,28: number analyzed (Participants) | 35 | 37 | 36 | 35 | 28 | 28
  CD3+CD4+ treg flow cyto;Week 4;n=35,37,36,35,28,28 | 0.0117 (0.2048) | 0.0575 (0.2571) | 0.0825 (0.1875) | 0.0135 (0.2167) | -0.0229 (0.2878) | 0.1215 (0.2442)
  CD3+CD4+ treg flow cyto;Week 8;n=31,35,32,36,27,25: number analyzed (Participants) | 31 | 35 | 32 | 36 | 27 | 25
  CD3+CD4+ treg flow cyto;Week 8;n=31,35,32,36,27,25 | 0.0286 (0.1744) | 0.0687 (0.2923) | -0.0158 (0.2536) | -0.0284 (0.2018) | -0.0007 (0.2751) | 0.0849 (0.1883)
  CD3+CD4+treg flow cyto;Week 12;n=32,36,31,32,25,24: number analyzed (Participants) | 32 | 36 | 31 | 32 | 25 | 24
  CD3+CD4+treg flow cyto;Week 12;n=32,36,31,32,25,24 | 0.0235 (0.2508) | 0.1058 (0.2718) | 0.0979 (0.2691) | 0.0141 (0.1885) | -0.0403 (0.3331) | 0.0213 (0.1940)
  CD16+CD56+; Week 4; n=37,38,38,37,29,32: number analyzed (Participants) | 37 | 38 | 38 | 37 | 29 | 32
  CD16+CD56+; Week 4; n=37,38,38,37,29,32 | -0.021 (0.0942) | -0.018 (0.0752) | -0.019 (0.0976) | -0.004 (0.1057) | -0.009 (0.0837) | 0.016 (0.0999)
  CD16+CD56+; Week 8; n=34,37,34,37,28,27: number analyzed (Participants) | 34 | 37 | 34 | 37 | 28 | 27
  CD16+CD56+; Week 8; n=34,37,34,37,28,27 | -0.013 (0.0909) | -0.012 (0.1594) | -0.016 (0.1045) | -0.009 (0.0919) | -0.029 (0.0860) | -0.012 (0.1131)
  CD16+CD56+; Week 12; n= 35,37,32,34,27,27: number analyzed (Participants) | 35 | 37 | 32 | 34 | 27 | 27
  CD16+CD56+; Week 12; n= 35,37,32,34,27,27 | -0.038 (0.0884) | -0.021 (0.0911) | -0.022 (0.0792) | -0.036 (0.0702) | -0.039 (0.0909) | -0.020 (0.0888)
  CD3+CD4+CD25+CD127; Week4;n=35,37,36,35,28,28: number analyzed (Participants) | 35 | 37 | 36 | 35 | 28 | 28
  CD3+CD4+CD25+CD127; Week4;n=35,37,36,35,28,28 | 0.0006 (0.0139) | 0.0023 (0.0150) | 0.0022 (0.0172) | 0.0005 (0.0174) | -0.0050 (0.0179) | 0.0098 (0.0345)
  CD3+CD4+CD25+CD127; Week8;n=31,35,32,36,27,25: number analyzed (Participants) | 31 | 35 | 32 | 36 | 27 | 25
  CD3+CD4+CD25+CD127; Week8;n=31,35,32,36,27,25 | 0.0044 (0.0199) | 0.0062 (0.0167) | 0.0026 (0.0223) | 0.0029 (0.0196) | -0.0049 (0.0181) | 0.0054 (0.0222)
  CD3+CD4+CD25+CD127; Week12;n=32,36,31,32,25,24: number analyzed (Participants) | 32 | 36 | 31 | 32 | 25 | 24
  CD3+CD4+CD25+CD127; Week12;n=32,36,31,32,25,24 | 0.0050 (0.0193) | 0.0056 (0.0228) | 0.0081 (0.0229) | 0.0054 (0.0217) | 0.0007 (0.0230) | 0.0055 (0.0215)
  CD3+CD4+foxP3+CD25+CD127;Week4;n=35,37,36,35,28,28: number analyzed (Participants) | 35 | 37 | 36 | 35 | 28 | 28
  CD3+CD4+foxP3+CD25+CD127;Week4;n=35,37,36,35,28,28 | 0.0009 (0.0125) | 0.0001 (0.0162) | 0.0009 (0.0129) | -0.0013 (0.0164) | 0.0008 (0.0099) | 0.0056 (0.0123)
  CD3+CD4+foxP3+CD25+CD127;Week8;n=31,35,32,35,27,25: number analyzed (Participants) | 31 | 35 | 32 | 35 | 27 | 25
  CD3+CD4+foxP3+CD25+CD127;Week8;n=31,35,32,35,27,25 | 0.0070 (0.0184) | 0.0011 (0.0147) | 0.0021 (0.0182) | -0.0015 (0.0151) | 0.0032 (0.0151) | 0.0047 (0.0166)
  CD3+CD4+foxP3+CD25+CD127Week12;n=32,36,31,32,25,24: number analyzed (Participants) | 32 | 36 | 31 | 32 | 25 | 24
  CD3+CD4+foxP3+CD25+CD127Week12;n=32,36,31,32,25,24 | 0.0076 (0.0149) | 0.0003 (0.0198) | 0.0052 (0.0192) | -0.0012 (0.0180) | 0.0039 (0.0160) | 0.0059 (0.0127)
  T &B cell NK lympho; Week4;n=37,38,38,37,29,32: number analyzed (Participants) | 37 | 38 | 38 | 37 | 29 | 32
  T &B cell NK lympho; Week4;n=37,38,38,37,29,32 | 0.009 (0.5461) | 0.101 (0.5287) | 0.092 (0.5122) | 0.021 (0.4664) | -0.082 (0.6206) | 0.228 (0.5116)
  T &B cell NK lympho;Week8;n=34,37,34,37,28,27: number analyzed (Participants) | 34 | 37 | 34 | 37 | 28 | 27
  T &B cell NK lympho;Week8;n=34,37,34,37,28,27 | 0.059 (0.4430) | 0.083 (0.6737) | 0.025 (0.5688) | -0.070 (0.4141) | -0.109 (0.6219) | 0.132 (0.5150)
  T &B cell NK lympho; Week12;n=35,37,32,34,27,27: number analyzed (Participants) | 35 | 37 | 32 | 34 | 27 | 27
  T &B cell NK lympho; Week12;n=35,37,32,34,27,27 | -0.041 (0.5922) | 0.174 (0.5825) | 0.140 (0.5609) | -0.009 (0.4041) | -0.236 (0.6830) | -0.001 (0.3842)

33. Secondary Outcome: Number of Participants With Immunopheotyping Data Outside the Reference Range
Description: Blood samples were collected from participants for evaluation of immunophenotyping parameters by Potential Clinical Importance Criteria at Baseline, Week 4, Week 8, Week 12 nd any visit post-screen. The immunophenotyping parameters included CD 19, CD3, CD3+CD8+, CD3+CD4+, CD16+CD56+, CD3+CD4+CD25+CD127, CD3+CD4+foxP3+CD25+CD127 and T and NK lympho. CD3, CD3+CD8+ and CD3+CD4+ were also evaluated by using treg flow cyto. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline, Week, 4, 8, 12 and post-screen (up to Week 16)
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  CD19; Baseline; n=40,41,43,40,41,40: number analyzed (Participants) | 40 | 41 | 43 | 40 | 41 | 40
  CD19; Baseline; n=40,41,43,40,41,40 | 0 | 0 | 5 | 2 | 1 | 2
  CD19; Week 4; n= 37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  CD19; Week 4; n= 37,38,38,38,30,32 | 3 | 0 | 5 | 4 | 1 | 2
  CD19; Week 8; n= 34,37,34,38,29,27: number analyzed (Participants) | 34 | 37 | 34 | 38 | 29 | 27
  CD19; Week 8; n= 34,37,34,38,29,27 | 2 | 1 | 3 | 4 | 3 | 2
  CD19; Week 12; n= 35,37,32,35,28,27: number analyzed (Participants) | 35 | 37 | 32 | 35 | 28 | 27
  CD19; Week 12; n= 35,37,32,35,28,27 | 1 | 3 | 3 | 3 | 0 | 1
  CD19; post-screen; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD19; post-screen; n= 38,39,38,39,30,32 | 4 | 3 | 7 | 7 | 3 | 4
  CD3; Baseline; n=40,41,43,41,41,40: number analyzed (Participants) | 40 | 41 | 43 | 41 | 41 | 40
  CD3; Baseline; n=40,41,43,41,41,40 | 8 | 3 | 6 | 1 | 4 | 3
  CD3; Week 4; n=37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  CD3; Week 4; n=37,38,38,38,30,32 | 6 | 3 | 6 | 2 | 4 | 1
  CD3; Week 8; n=34,37,34,38,29,27: number analyzed (Participants) | 34 | 37 | 34 | 38 | 29 | 27
  CD3; Week 8; n=34,37,34,38,29,27 | 5 | 3 | 5 | 2 | 2 | 4
  CD3; Week 12; n=35,37,32,35,28,27: number analyzed (Participants) | 35 | 37 | 32 | 35 | 28 | 27
  CD3; Week 12; n=35,37,32,35,28,27 | 4 | 2 | 5 | 1 | 2 | 2
  CD3; post-screen; n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3; post-screen; n=38,39,38,39,30,32 | 8 | 5 | 9 | 4 | 6 | 7
  CD3 treg flow cyto;Baseline; n=38,40,42,39,40,37: number analyzed (Participants) | 38 | 40 | 42 | 39 | 40 | 37
  CD3 treg flow cyto;Baseline; n=38,40,42,39,40,37 | 0 | 0 | 0 | 0 | 0 | 0
  CD3 treg flow cyto; Week 4; n=37,38,37,37,30,30: number analyzed (Participants) | 37 | 38 | 37 | 37 | 30 | 30
  CD3 treg flow cyto; Week 4; n=37,38,37,37,30,30 | 0 | 0 | 0 | 0 | 0 | 0
  CD3 treg flow cyto; Week8; n=33,36,33,38,29,26: number analyzed (Participants) | 33 | 36 | 33 | 38 | 29 | 26
  CD3 treg flow cyto; Week8; n=33,36,33,38,29,26 | 0 | 0 | 0 | 0 | 0 | 0
  CD3 treg flow cyto; Week 12; n= 34,37,32,34,27,25: number analyzed (Participants) | 34 | 37 | 32 | 34 | 27 | 25
  CD3 treg flow cyto; Week 12; n= 34,37,32,34,27,25 | 0 | 0 | 1 | 0 | 0 | 0
  CD3treg flow cyto; postscreen; n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3treg flow cyto; postscreen; n=38,39,38,39,30,32 | 0 | 0 | 1 | 0 | 0 | 0
  CD3+CD8+; Baseline; n= 40,41,43,40,41,40: number analyzed (Participants) | 40 | 41 | 43 | 40 | 41 | 40
  CD3+CD8+; Baseline; n= 40,41,43,40,41,40 | 9 | 3 | 3 | 2 | 5 | 4
  CD3+CD8+; Week 4; n=37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  CD3+CD8+; Week 4; n=37,38,38,38,30,32 | 5 | 3 | 4 | 3 | 3 | 3
  CD3+CD8+; Week 8; n=34,37,34,38,29,27: number analyzed (Participants) | 34 | 37 | 34 | 38 | 29 | 27
  CD3+CD8+; Week 8; n=34,37,34,38,29,27 | 4 | 2 | 4 | 2 | 1 | 3
  CD3+CD8+; Week 12; n= 35,37,32,35,28,27: number analyzed (Participants) | 35 | 37 | 32 | 35 | 28 | 27
  CD3+CD8+; Week 12; n= 35,37,32,35,28,27 | 3 | 3 | 4 | 1 | 1 | 4
  CD3+CD8+; post-screen; n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3+CD8+; post-screen; n=38,39,38,39,30,32 | 8 | 4 | 8 | 4 | 5 | 6
  CD3+CD8+tregflowcyto;Baseline;n= 38,40,42,39,40,37: number analyzed (Participants) | 38 | 40 | 42 | 39 | 40 | 37
  CD3+CD8+tregflowcyto;Baseline;n= 38,40,42,39,40,37 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD8+tregflowcyto;Week4;n=37,38,37,37,30,30: number analyzed (Participants) | 37 | 38 | 37 | 37 | 30 | 30
  CD3+CD8+tregflowcyto;Week4;n=37,38,37,37,30,30 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD8+tregflowcyto;Week8;n=33,36,33,38,29,26: number analyzed (Participants) | 33 | 36 | 33 | 38 | 29 | 26
  CD3+CD8+tregflowcyto;Week8;n=33,36,33,38,29,26 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD8+tregflowcyto;Week12;n=34,37,32,34,27,25: number analyzed (Participants) | 34 | 37 | 32 | 34 | 27 | 25
  CD3+CD8+tregflowcyto;Week12;n=34,37,32,34,27,25 | 0 | 0 | 1 | 0 | 0 | 0
  CD3+CD8+tregflowcytopostscreen;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3+CD8+tregflowcytopostscreen;n=38,39,38,39,30,32 | 0 | 0 | 1 | 0 | 0 | 0
  CD3+CD4+; Baseline;n=40,41,43,40,41,40: number analyzed (Participants) | 40 | 41 | 43 | 40 | 41 | 40
  CD3+CD4+; Baseline;n=40,41,43,40,41,40 | 8 | 5 | 6 | 3 | 4 | 2
  CD3+CD4+; Week 4; n=37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  CD3+CD4+; Week 4; n=37,38,38,38,30,32 | 5 | 4 | 3 | 3 | 3 | 1
  CD3+CD4+; Week 8; n=34,37,34,38,29,27: number analyzed (Participants) | 34 | 37 | 34 | 38 | 29 | 27
  CD3+CD4+; Week 8; n=34,37,34,38,29,27 | 4 | 6 | 3 | 5 | 6 | 3
  CD3+CD4+; Week 12; n= 35,37,32,35,28,27: number analyzed (Participants) | 35 | 37 | 32 | 35 | 28 | 27
  CD3+CD4+; Week 12; n= 35,37,32,35,28,27 | 5 | 6 | 5 | 2 | 7 | 4
  CD3+CD4+; post-screen;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3+CD4+; post-screen;n=38,39,38,39,30,32 | 8 | 8 | 7 | 7 | 9 | 7
  CD3+CD4+tregflow cyto;Baseline;n=38,40,42,39,40,37: number analyzed (Participants) | 38 | 40 | 42 | 39 | 40 | 37
  CD3+CD4+tregflow cyto;Baseline;n=38,40,42,39,40,37 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+tregflow cyto;Week4;n=37,38,37,37, 30,30: number analyzed (Participants) | 37 | 38 | 37 | 37 | 30 | 30
  CD3+CD4+tregflow cyto;Week4;n=37,38,37,37, 30,30 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+tregflow cyto;Week8;n=33,36,33,38,29,26: number analyzed (Participants) | 33 | 36 | 33 | 38 | 29 | 26
  CD3+CD4+tregflow cyto;Week8;n=33,36,33,38,29,26 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+tregflow cyto;Week12;n=34,37,32,34,27,25: number analyzed (Participants) | 34 | 37 | 32 | 34 | 27 | 25
  CD3+CD4+tregflow cyto;Week12;n=34,37,32,34,27,25 | 0 | 0 | 1 | 0 | 0 | 0
  CD3+CD4+tregflow;postscreen;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3+CD4+tregflow;postscreen;n=38,39,38,39,30,32 | 0 | 0 | 1 | 0 | 0 | 0
  CD16+CD56+;Baseline;n=40,41,43,40,41,40: number analyzed (Participants) | 40 | 41 | 43 | 40 | 41 | 40
  CD16+CD56+;Baseline;n=40,41,43,40,41,40 | 1 | 1 | 2 | 1 | 1 | 0
  CD16+CD56+;Week4;n=37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  CD16+CD56+;Week4;n=37,38,38,38,30,32 | 0 | 0 | 1 | 1 | 1 | 1
  CD16+CD56+;Week8;n=34,37,34,38,29,27: number analyzed (Participants) | 34 | 37 | 34 | 38 | 29 | 27
  CD16+CD56+;Week8;n=34,37,34,38,29,27 | 1 | 2 | 1 | 0 | 0 | 1
  CD16+CD56+;Week12;n=35,37,32,35,28,27: number analyzed (Participants) | 35 | 37 | 32 | 35 | 28 | 27
  CD16+CD56+;Week12;n=35,37,32,35,28,27 | 0 | 0 | 3 | 0 | 0 | 0
  CD16+CD56+;postscreen;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD16+CD56+;postscreen;n=38,39,38,39,30,32 | 1 | 2 | 3 | 1 | 1 | 1
  CD3+CD4+CD25+CD127;Baseline;n=38,40,42,39,40,37: number analyzed (Participants) | 38 | 40 | 42 | 39 | 40 | 37
  CD3+CD4+CD25+CD127;Baseline;n=38,40,42,39,40,37 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+CD25+CD127;Week 4;n=37,38,37,37,30,30: number analyzed (Participants) | 37 | 38 | 37 | 37 | 30 | 30
  CD3+CD4+CD25+CD127;Week 4;n=37,38,37,37,30,30 | 3 | 2 | 1 | 3 | 4 | 1
  CD3+CD4+CD25+CD127;Week8;n=33,36,33,38,29,26: number analyzed (Participants) | 33 | 36 | 33 | 38 | 29 | 26
  CD3+CD4+CD25+CD127;Week8;n=33,36,33,38,29,26 | 4 | 3 | 3 | 6 | 2 | 4
  CD3+CD4+CD25+CD127;Week12;n=34,37,32,34,27,25: number analyzed (Participants) | 34 | 37 | 32 | 34 | 27 | 25
  CD3+CD4+CD25+CD127;Week12;n=34,37,32,34,27,25 | 4 | 4 | 6 | 6 | 5 | 5
  CD3+CD4+CD25+CD127;postscreen;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3+CD4+CD25+CD127;postscreen;n=38,39,38,39,30,32 | 7 | 6 | 8 | 9 | 9 | 7
  CD3+CD4+foxP3+CD25+CD127;Base;n=38,40,42,39,40,37: number analyzed (Participants) | 38 | 40 | 42 | 39 | 40 | 37
  CD3+CD4+foxP3+CD25+CD127;Base;n=38,40,42,39,40,37 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+foxP3+CD25+CD127;Week4;n=37,38,37,37,30,30: number analyzed (Participants) | 37 | 38 | 37 | 37 | 30 | 30
  CD3+CD4+foxP3+CD25+CD127;Week4;n=37,38,37,37,30,30 | 10 | 10 | 7 | 11 | 6 | 7
  CD3+CD4+foxP3+CD25+CD127;Week8;n=33,36,33,37,29,26: number analyzed (Participants) | 33 | 36 | 33 | 37 | 29 | 26
  CD3+CD4+foxP3+CD25+CD127;Week8;n=33,36,33,37,29,26 | 9 | 8 | 14 | 9 | 6 | 9
  CD3+CD4+foxP3+CD25+CD127;Week12;34,37,32,34,27,25: number analyzed (Participants) | 34 | 37 | 32 | 34 | 27 | 25
  CD3+CD4+foxP3+CD25+CD127;Week12;34,37,32,34,27,25 | 10 | 9 | 9 | 14 | 8 | 6
  CD3+CD4+foxP3+CD25+CD127;post;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  CD3+CD4+foxP3+CD25+CD127;post;n=38,39,38,39,30,32 | 19 | 19 | 21 | 22 | 16 | 13
  T-B cell NK lympho;Baseline; n=40,41,43,40,41,40: number analyzed (Participants) | 40 | 41 | 43 | 40 | 41 | 40
  T-B cell NK lympho;Baseline; n=40,41,43,40,41,40 | 1 | 1 | 2 | 0 | 0 | 1
  T-B cell NK lympho;Week4; n=37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  T-B cell NK lympho;Week4; n=37,38,38,38,30,32 | 0 | 1 | 0 | 0 | 2 | 0
  T-B cell NK lympho;Week8;n=34,37,34,38,29,27: number analyzed (Participants) | 34 | 37 | 34 | 38 | 29 | 27
  T-B cell NK lympho;Week8;n=34,37,34,38,29,27 | 0 | 1 | 1 | 2 | 0 | 0
  T-B cell NK lympho;Week12;n=35,37,32,35,28,27: number analyzed (Participants) | 35 | 37 | 32 | 35 | 28 | 27
  T-B cell NK lympho;Week12;n=35,37,32,35,28,27 | 0 | 0 | 1 | 0 | 3 | 0
  T-B cell NK lympho;postscreen;n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  T-B cell NK lympho;postscreen;n=38,39,38,39,30,32 | 0 | 1 | 2 | 2 | 5 | 0

34. Secondary Outcome: Change From Baseline in Immunoglobin (Ig) A, IgG and IgM Levels
Description: Blood samples were collected to evaluate change from Baseline in IgA, IgG, IM values at Baseline throughout the 12 weeks of study treatment. Baseline values were taken at Day 1 and change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week, 4, 8 and 12
Population: Safety population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
G/L
  IgA; Week 4; n= 37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  IgA; Week 4; n= 37,38,38,38,30,32 | -0.016 (0.2528) | -0.103 (0.2108) | -0.079 (0.2003) | -0.026 (0.2342) | -0.046 (0.2179) | -0.045 (0.3141)
  IgA; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  IgA; Week 8; n= 35,37,34,38,29,28 | -0.064 (0.2558) | -0.116 (0.2314) | -0.056 (0.2570) | 0.035 (0.2188) | 0.026 (0.2695) | -0.036 (0.3106)
  IgA; Week 12; n= 36,37,32,35,28,27: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 27
  IgA; Week 12; n= 36,37,32,35,28,27 | -0.056 (0.2820) | -0.099 (0.6148) | -0.140 (0.2207) | -0.042 (0.2657) | -0.038 (0.1744) | -0.016 (0.2462)
  IgG; Week 4; n= 37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  IgG; Week 4; n= 37,38,38,38,30,32 | -0.130 (1.0945) | -0.446 (0.8854) | -0.282 (1.2618) | -0.347 (1.1148) | -0.198 (1.2753) | -0.112 (1.1564)
  IgG; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  IgG; Week 8; n= 35,37,34,38,29,28 | -0.007 (1.2785) | -0.457 (1.0787) | -0.121 (1.4233) | -0.200 (1.1449) | 0.428 (1.1984) | 0.203 (1.4037)
  IgG; Week 12; n= 36,37,32,35,28,27: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 27
  IgG; Week 12; n= 36,37,32,35,28,27 | -0.033 (1.2978) | -0.436 (3.8561) | -0.367 (1.0214) | -0.269 (0.9239) | 0.256 (1.5915) | 0.331 (0.8796)
  IgM; Week 4; n=37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  IgM; Week 4; n=37,38,38,38,30,32 | -0.049 (0.1524) | -0.102 (0.1514) | -0.077 (0.0968) | -0.043 (0.1303) | -0.052 (0.0933) | -0.040 (0.0886)
  IgM; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  IgM; Week 8; n= 35,37,34,38,29,28 | -0.070 (0.1069) | -0.095 (0.1314) | -0.111 (0.1290) | -0.052 (0.1167) | -0.014 (0.1396) | -0.040 (0.0956)
  IgM; Week 12; n= 36,37,32,35,28,27: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 27
  IgM; Week 12; n= 36,37,32,35,28,27 | -0.055 (0.1852) | -0.098 (0.1955) | -0.125 (0.1233) | -0.072 (0.1112) | -0.047 (0.1300) | -0.034 (0.0850)

35. Secondary Outcome: Number of Participants With Immunoglobulin Data Outside the Reference Range
Description: Blood samples were collected from participants for evaluation of immunoglobulin data outside the reference range at Baseline, Week 4, Week 8, Week 12 and any visit post-screen. The immunoglobulin parameters included IgA, IgG and Ig M. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline, Week, 4, 8, 12, post-screen (up to Week 16)
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  IgA; Baseline; n= 40,41,43,41,42,40 | 2 | 3 | 2 | 1 | 4 | 2
  IgA; Week 4; n= 37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  IgA; Week 4; n= 37,38,38,38,30,32 | 2 | 2 | 3 | 0 | 3 | 2
  IgA; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  IgA; Week 8; n= 35,37,34,38,29,28 | 2 | 1 | 3 | 2 | 1 | 2
  IgA; Week 12; n= 36,37,32,35,28,27: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 27
  IgA; Week 12; n= 36,37,32,35,28,27 | 3 | 1 | 4 | 1 | 1 | 2
  IgA; post-screen; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  IgA; post-screen; n= 38,39,38,39,30,32 | 4 | 3 | 4 | 2 | 3 | 3
  IgG; Baseline; n=40,41,43,41,42,40 | 2 | 5 | 1 | 4 | 3 | 3
  IgG; Week 4; n= 37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  IgG; Week 4; n= 37,38,38,38,30,32 | 1 | 3 | 0 | 3 | 3 | 2
  IgG; Week 8; n=35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  IgG; Week 8; n=35,37,34,38,29,28 | 3 | 3 | 0 | 3 | 4 | 2
  IgG; Week 12; n=36,37,32,35,28,27: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 27
  IgG; Week 12; n=36,37,32,35,28,27 | 4 | 5 | 0 | 5 | 4 | 2
  IgG; post screen; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  IgG; post screen; n= 38,39,38,39,30,32 | 4 | 6 | 0 | 5 | 6 | 3
  IgM;Baseline; n= 40,41,43,41,42,40 | 4 | 7 | 3 | 3 | 6 | 4
  IgM; Week 4; n=37,38,38,38,30,32: number analyzed (Participants) | 37 | 38 | 38 | 38 | 30 | 32
  IgM; Week 4; n=37,38,38,38,30,32 | 3 | 5 | 6 | 1 | 2 | 6
  IgM; Week 8; n= 35,37,34,38,29,28: number analyzed (Participants) | 35 | 37 | 34 | 38 | 29 | 28
  IgM; Week 8; n= 35,37,34,38,29,28 | 3 | 4 | 7 | 3 | 3 | 5
  IgM; Week12; n= 36,37,32,35,28,27: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 27
  IgM; Week12; n= 36,37,32,35,28,27 | 4 | 5 | 7 | 2 | 3 | 6
  IgM; post-screen; n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  IgM; post-screen; n=38,39,38,39,30,32 | 4 | 5 | 10 | 4 | 3 | 6

36. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured from Baseline up to follow up Visit 1 at Week 14 in semi-supine position after at least 5 minutes of rest. The Baseline value was taken at Day 1 and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 1, 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Millimeter of mercury (mmHg)
  SBP; Week 1; n= 38,31,39,37,38,33: number analyzed (Participants) | 38 | 31 | 39 | 37 | 38 | 33
  SBP; Week 1; n= 38,31,39,37,38,33 | -1.6 (8.89) | -2.3 (11.02) | -2.3 (14.72) | -1.9 (9.77) | 0.8 (9.32) | -0.7 (9.45)
  SBP; Week 2; n=39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  SBP; Week 2; n=39,39,39,39,33,32 | -1.7 (12.22) | 0.6 (10.57) | -4.3 (13.37) | -1.2 (11.41) | -0.8 (10.41) | -1.6 (6.90)
  SBP; Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  SBP; Week 4; n= 38,39,38,39,30,32 | -1.7 (10.57) | 0.5 (10.00) | -3.8 (9.05) | -1.8 (11.94) | 1.9 (13.33) | -0.5 (14.24)
  SBP; Week 8; n= 36,37,34,38,29,28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  SBP; Week 8; n= 36,37,34,38,29,28 | -1.9 (10.74) | -0.5 (11.27) | -4.3 (11.38) | -1.9 (9.86) | 0.0 (11.29) | 1.0 (17.08)
  SBP; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  SBP; Week 12; n= 36,37,32,35,28,28 | -3.1 (10.28) | -0.1 (11.64) | -1.9 (12.62) | -2.4 (10.71) | -0.5 (10.44) | -0.5 (12.67)
  SBP; Week 14; n=34,35,32,34,31,29: number analyzed (Participants) | 34 | 35 | 32 | 34 | 31 | 29
  SBP; Week 14; n=34,35,32,34,31,29 | -1.0 (11.95) | -0.5 (12.52) | -1.4 (12.76) | -1.9 (9.46) | 1.2 (13.18) | 0.3 (11.29)
  SBP; EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  SBP; EW; n= 3,4,7,3,11,11 | 5.3 (8.08) | -5.3 (18.01) | 4.9 (13.63) | -0.7 (7.37) | 1.2 (8.81) | 2.0 (6.96)
  DBP; Week 1; n=38,31,39,37,38,33: number analyzed (Participants) | 38 | 31 | 39 | 37 | 38 | 33
  DBP; Week 1; n=38,31,39,37,38,33 | -2.0 (8.55) | 1.4 (8.48) | -1.9 (8.74) | -1.5 (7.33) | 1.1 (9.29) | -0.4 (7.53)
  DBP; Week 2; n=39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  DBP; Week 2; n=39,39,39,39,33,32 | -3.4 (9.60) | 0.1 (8.14) | -3.7 (7.63) | -3.3 (7.07) | -2.2 (10.29) | -0.9 (5.97)
  DBP; Week 4; n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  DBP; Week 4; n=38,39,38,39,30,32 | -3.0 (12.21) | 0.9 (7.98) | -3.1 (9.31) | -4.0 (7.98) | -0.1 (10.49) | 1.9 (9.18)
  DBP; Week 8; n=36,37,34,38,29,28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  DBP; Week 8; n=36,37,34,38,29,28 | -4.8 (9.79) | 1.0 (8.07) | -3.3 (9.24) | -2.1 (8.91) | -0.2 (10.10) | 2.2 (10.08)
  DBP; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  DBP; Week 12; n= 36,37,32,35,28,28 | -6.5 (8.86) | 2.6 (7.02) | -2.8 (8.82) | -4.0 (9.18) | 0.9 (9.81) | 1.3 (8.93)
  DBP; Week 14; n= 34,35,32,34,31,29: number analyzed (Participants) | 34 | 35 | 32 | 34 | 31 | 29
  DBP; Week 14; n= 34,35,32,34,31,29 | -5.6 (9.23) | -0.5 (7.71) | -2.9 (9.10) | -0.4 (8.49) | -0.4 (9.45) | 0.9 (7.75)
  DBP; EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  DBP; EW; n= 3,4,7,3,11,11 | 3.3 (3.06) | 1.3 (3.40) | 0.0 (10.82) | -1.0 (9.54) | 2.3 (3.66) | -2.7 (7.02)

37. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate were measured from Baseline up to follow up Visit 1 at Week 14 in semi-supine position after at least 5 minutes of rest. The Baseline value was taken at Day 1 and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 1, 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Beats per minute (bpm)
  Week 1; n= 38,41,39,37,38,33: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 33
  Week 1; n= 38,41,39,37,38,33 | 5.8 (9.19) | 2.5 (8.68) | 0.8 (10.19) | -0.4 (9.39) | 0.4 (9.43) | -0.4 (9.82)
  Week 2; n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Week 2; n= 39,39,39,39,33,32 | 3.7 (10.67) | 2.3 (10.90) | 0.1 (9.63) | 1.0 (10.90) | 1.5 (11.99) | 1.0 (10.47)
  Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38,39,38,39,30,32 | 6.2 (10.02) | 0.6 (10.79) | -0.3 (12.30) | 0.4 (10.88) | -1.7 (11.67) | 0.1 (8.42)
  Week 8; n= 36,37,34,38,29,28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Week 8; n= 36,37,34,38,29,28 | 4.1 (9.72) | 0.6 (10.27) | -1.7 (9.59) | 3.2 (11.23) | -0.2 (11.45) | 0.8 (8.97)
  Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; n= 36,37,32,35,28,28 | 3.0 (10.03) | -0.0 (11.55) | 0.0 (10.08) | 0.4 (9.74) | -1.9 (9.58) | 1.3 (10.76)
  Week 14; n= 34,35,32,34,31,29: number analyzed (Participants) | 34 | 35 | 32 | 34 | 31 | 29
  Week 14; n= 34,35,32,34,31,29 | 3.3 (9.38) | 3.5 (11.65) | 0.6 (10.00) | 2.5 (10.97) | 0.8 (11.06) | 0.7 (8.56)
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | -13.7 (1.15) | 0.3 (3.50) | -6.0 (9.83) | -2.7 (8.96) | 4.2 (12.18) | -0.5 (9.15)

38. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature were measured from Baseline up to follow up Visit 1 at Week 14 in semi-supine position after at least 5 minutes of rest. The Baseline value was taken at Day 1 and change from Baseline was defined as post dose visit value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were measured.
Time Frame: Week 1, 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Degree Celsius
  Week 1; n= 38,41,39, 37,38,33: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 33
  Week 1; n= 38,41,39, 37,38,33 | 0.013 (0.3640) | -0.056 (0.2618) | 0.015 (0.3689) | -0.006 (0.3932) | -0.053 (0.7928) | -0.024 (0.2693)
  Week 2; n=39,39,39,39,32,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 32 | 32
  Week 2; n=39,39,39,39,32,32 | -0.054 (0.4973) | -0.064 (0.2680) | 0.005 (0.3332) | -0.069 (0.4691) | -0.097 (0.7082) | 0.016 (0.2841)
  Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Week 4; n= 38,39,38,39,30,32 | -0.074 (0.4428) | -0.023 (0.3256) | -0.013 (0.3458) | -0.068 (0.4902) | -0.030 (0.6706) | 0.013 (0.2459)
  Week 8; n= 36,37,34,38,29,28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Week 8; n= 36,37,34,38,29,28 | 0.006 (0.4276) | -0.024 (0.2671) | -0.056 (0.3295) | 0.045 (0.4011) | 0.062 (0.7566) | 0.021 (0.3304)
  Week 12; n=36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; n=36,37,32,35,28,28 | 0.003 (0.4212) | -0.068 (0.3292) | -0.078 (0.2814) | -0.040 (0.4532) | 0.043 (0.7618) | 0.004 (0.4574)
  Week 14;n=34,35,32,34,31,29: number analyzed (Participants) | 34 | 35 | 32 | 34 | 31 | 29
  Week 14;n=34,35,32,34,31,29 | -0.079 (0.4059) | -0.131 (0.6416) | -0.059 (0.3618) | -0.109 (0.4876) | -0.013 (0.8740) | -0.052 (0.3582)
  EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  EW; n= 3,4,7,3,11,11 | -0.033 (0.1528) | 0.000 (0.3651) | 0.100 (0.2517) | 0.400 (0.5568) | -0.182 (0.5212) | 0.164 (0.4985)

39. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Blood samples were collected from participants for evaluation of vital signs by Potential Clinical Importance Criteria from Baseline to Week 14, EW and any visit post-screen. The vital signs included SBP, DBP and pulse rate. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline, Week 2, 4, 8, 12, 14, EW (up to week 14)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  SBP; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 1
  SBP; Week 1; n= 38,41,39,37,38,33: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 33
  SBP; Week 1; n= 38,41,39,37,38,33 | 1 | 1 | 0 | 0 | 0 | 0
  SBP; Week 2; n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  SBP; Week 2; n= 39,39,39,39,33,32 | 0 | 0 | 0 | 2 | 0 | 1
  SBP; Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  SBP; Week 4; n= 38,39,38,39,30,32 | 0 | 0 | 0 | 1 | 0 | 1
  SBP; Week 8; n= 36,37,34,38,29,28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  SBP; Week 8; n= 36,37,34,38,29,28 | 0 | 0 | 0 | 0 | 0 | 2
  SBP; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  SBP; Week 12; n= 36,37,32,35,28,28 | 0 | 1 | 1 | 1 | 0 | 1
  SBP: Week 14; n= 34,35,32,34,31,29: number analyzed (Participants) | 34 | 35 | 32 | 34 | 31 | 29
  SBP: Week 14; n= 34,35,32,34,31,29 | 0 | 0 | 0 | 2 | 0 | 1
  SBP; EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  SBP; EW; n= 3,4,7,3,11,11 | 0 | 0 | 0 | 0 | 0 | 0
  SBP; post-screen; n= 40,41,43,41,42,40 | 1 | 2 | 1 | 3 | 0 | 3
  DBP; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 1 | 0 | 0 | 0
  DBP; Week 1; n=38,41,39,37,38,33: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 33
  DBP; Week 1; n=38,41,39,37,38,33 | 0 | 0 | 0 | 0 | 0 | 0
  DBP; Week 2; n=39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  DBP; Week 2; n=39,39,39,39,33,32 | 0 | 0 | 0 | 0 | 1 | 0
  DBP; Week 4; n=38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  DBP; Week 4; n=38,39,38,39,30,32 | 0 | 0 | 0 | 0 | 0 | 1
  DBP; Week 8; n= 36,37,34,38,29,28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  DBP; Week 8; n= 36,37,34,38,29,28 | 0 | 0 | 0 | 1 | 1 | 1
  DBP; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  DBP; Week 12; n= 36,37,32,35,28,28 | 0 | 0 | 0 | 1 | 1 | 0
  DBP; Week 14; n= 34,35,32,34,31,29: number analyzed (Participants) | 34 | 35 | 32 | 34 | 31 | 29
  DBP; Week 14; n= 34,35,32,34,31,29 | 0 | 0 | 0 | 1 | 0 | 0
  DBP; EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  DBP; EW; n= 3,4,7,3,11,11 | 1 | 0 | 0 | 0 | 0 | 0
  DBP; post-screen; n= 40,41,43,41,42,40 | 1 | 0 | 1 | 1 | 1 | 2
  Pulse rate; Baseline; n= 40,41,43,41,42,40 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate; Week 1; n= 38,41,39,37,38,33: number analyzed (Participants) | 38 | 41 | 39 | 37 | 38 | 33
  Pulse rate; Week 1; n= 38,41,39,37,38,33 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate;Week 2; n= 39,39,39,39,33,32: number analyzed (Participants) | 39 | 39 | 39 | 39 | 33 | 32
  Pulse rate;Week 2; n= 39,39,39,39,33,32 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate; Week 4; n= 38,39,38,39,30,32: number analyzed (Participants) | 38 | 39 | 38 | 39 | 30 | 32
  Pulse rate; Week 4; n= 38,39,38,39,30,32 | 0 | 0 | 0 | 1 | 0 | 0
  Pulse rate; Week 8; n= 36,37,34,38,29,28: number analyzed (Participants) | 36 | 37 | 34 | 38 | 29 | 28
  Pulse rate; Week 8; n= 36,37,34,38,29,28 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate; Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Pulse rate; Week 12; n= 36,37,32,35,28,28 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate; Week 14; n= 34,35,32,34,31,29: number analyzed (Participants) | 34 | 35 | 32 | 35 | 31 | 29
  Pulse rate; Week 14; n= 34,35,32,34,31,29 | 0 | 1 | 1 | 0 | 0 | 0
  Pulse rate; EW; n= 3,4,7,3,11,11: number analyzed (Participants) | 3 | 4 | 7 | 3 | 11 | 11
  Pulse rate; EW; n= 3,4,7,3,11,11 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate; post-screen; n=40,41,43,41,42,40 | 0 | 1 | 1 | 1 | 0 | 0

40. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single measurements of 12-lead ECGs were obtained at Baseline , Week 1, Week 12, Week 14 (follow up 1), EW and at any time post-screen using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc). Baseline was defined as the latest assessment prior to the first dose. For multiple ECGs at one visit, or "Any visit post-screen", a participant was categorized as "Abnormal" if >=1 assessment was abnormal. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline, Week 1, 12, 14, EW ( up to Week 14), post-screen
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 40 | 41 | 43 | 41 | 42 | 40
Participants
  Baseline; n= 40,41,43,41,42,40 | 8 | 6 | 4 | 5 | 5 | 5
  Week 1; n= 37,41,39,37,38,33: number analyzed (Participants) | 37 | 41 | 39 | 37 | 38 | 33
  Week 1; n= 37,41,39,37,38,33 | 8 | 8 | 4 | 5 | 5 | 6
  Week 12; n= 36,37,32,35,28,28: number analyzed (Participants) | 36 | 37 | 32 | 35 | 28 | 28
  Week 12; n= 36,37,32,35,28,28 | 7 | 6 | 4 | 3 | 1 | 4
  Week 14; n= 34,34,32,34,31,29: number analyzed (Participants) | 34 | 34 | 32 | 34 | 31 | 29
  Week 14; n= 34,34,32,34,31,29 | 8 | 4 | 5 | 6 | 1 | 5
  EW; n= 3,3,7,3,10,11: number analyzed (Participants) | 3 | 3 | 7 | 3 | 10 | 11
  EW; n= 3,3,7,3,10,11 | 0 | 1 | 0 | 2 | 0 | 1
  post-screen; n= 40,41,41,39,41,40: number analyzed (Participants) | 40 | 41 | 41 | 39 | 41 | 40
  post-screen; n= 40,41,41,39,41,40 | 12 | 10 | 5 | 8 | 5 | 9

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the Folow up Visit 2 at Week 16.
Description: AEs and SAEs were collected in Safety Population which comprised of all participants who received at least one dose of study treatment.
Arm/Group | GSK2894512 1% Cream Twice Daily | GSK2894512 1% Cream Once Daily | GSK2894512 0.5% Cream Twice Daily | GSK2894512 0.5% Cream Once Daily | Vehicle Cream Twice Daily | Vehicle Cream Once Daily
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41 | 0/43 | 0/41 | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/41 | 0/43 | 0/41 | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 28/40 | 22/41 | 20/43 | 23/41 | 19/42 | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2894512 1% Cream Twice Daily (N=40) | GSK2894512 1% Cream Once Daily (N=41) | GSK2894512 0.5% Cream Twice Daily (N=43) | GSK2894512 0.5% Cream Once Daily (N=41) | Vehicle Cream Twice Daily (N=42) | Vehicle Cream Once Daily (N=40)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit /hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2894512 1% Cream Twice Daily (N=40) | GSK2894512 1% Cream Once Daily (N=41) | GSK2894512 0.5% Cream Twice Daily (N=43) | GSK2894512 0.5% Cream Once Daily (N=41) | Vehicle Cream Twice Daily (N=42) | Vehicle Cream Once Daily (N=40)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (6) | 4 (5) | 1 (1) | 4 (4) | 3 (5)
Folliculitis (Infections and infestations) | 4 (4) | 8 (8) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory (Infections and infestations) | 4 (5) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema impetiginous (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sycosis barbae (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis follicularis et parafollicularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Application site reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye ulcer (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.